#### ViiV Healthcare group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for ING200336: A Prospective, Interventional Pharmacokinetic and Safety Study of DTG/ABC/3TC in Pregnant Women |
|---|---|---|
| <b>Compound Number</b> | : | GSK1349572+GR109714+GI265235 (GSK2619619) |
| Clinical Study<br>Identifier | : | ING200336 |
| Effective Date | : | 05-OCT-2021 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 200336.
- This RAP is intended to describe all the planned analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverables.
- The purpose of RAP Amendment 01 (to the originally approved RAP dated 03-MAR-2021) is to provide details on the Final (End of Study) analysis.

#### RAP Author(s):

| Author | Date |
|------------------------------------|-------------|
| Lead | |
| PPD | |
| Junior Statistician, Biostatistics | 04-OCT-2021 |
| Lead Statistician, Biostatistics | |

Copyright 2021 ViiV Healthcare group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **RAP Team Reviews:**

## **RAP Team Review Confirmations**

(Method: E-mail)

| Reviewer | Date |
|---|---|
| PPD | 04-OCT-2021 |
| Principal Statistician, Biostatistics, GSK | |
| PPD | 01-OCT-2021 |
| Principal Programmer/ Analyst, Biostatistics, GSK | 01 001 2021 |
| PPD | |
| PPD , ViiV | 03-OCT-2021 |
| PPD | |
| , Safety and Medical Governance, GSK | 04-OCT-2021 |
| PPD | 0.4.0.077.2021 |
| Clinical Development Leader, ViiV 04-OCT-2021 | |
| PPD | 04 OCT 2021 |
| Clinical Data Analyst, GSK | |
| PPD | 04 OCT 2021 |
| Manager- Statistics, Dev Biostats India Stats, GSK 04-OCT-2021 | |

# **Clinical Statistics and Clinical Programming Line Approvals:**

## Approved through email by:

| Approver | | | Date |
|---|---|---|---|
| Principal Statistician, Biostatistics, GSK | | 05-OCT-2021 | |
| PPD<br>PPD | Programming | | 05-OCT-2021 |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | DDUCTION | 6 |
| 2. | SUMM | IARY OF KEY PROTOCOL INFORMATION | 6 |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objectives and Endpoints | |
| | | 2.2.1. Study Design | |
| | 2.3. | Statistical Hypotheses / Statistical Analyses | 9 |
| | 2.4. | Interim Analyses | |
| | 2.5. | Final Analyses | 9 |
| 3. | ANALY | YSIS POPULATIONS | 10 |
| | 3.1. | Protocol Deviations | |
| 4. | | IDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | ENTIONS | |
| | 4.1. | Study Treatment & Sub-group Display Descriptors | |
| | 4.2. | Baseline Definitions | |
| | 4.3. | Multicentre Studies | |
| | 4.4. | Examination of Covariates, Other Strata and Subgroups | 11 |
| | 4.5. | Other Considerations for Data Analyses and Data Handling Conventions | 11 |
| 5. | | Y POPULATION ANALYSES | |
| | 5.1. | Overview of Planned Study Population Analyses | 13 |
| 6. | EFFIC | ACY ANALYSES | 15 |
| | 6.1. | Endpoint / Variables | 15 |
| | 6.2. | Summary Measure | |
| | 6.3. | Population of Interest | |
| | 6.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | 6.5. | Efficacy Analyses / Methods | 15 |
| 7. | SAFET | TY ANALYSES | 17 |
| | 7.1. | Adverse Events Analyses | 17 |
| | 7.2. | Clinical Laboratory and Other Safety Analyses | |
| 8. | рнурі | MACOKINETIC ANALYSES | 20 |
| 0. | 8.1. | Primary and Secondary Pharmacokinetic Analyses | |
| | 0.1. | 8.1.1. Endpoint / Variables | |
| | | 8.1.1.1. Drug Concentration Measures | |
| | | 8.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 8.1.2. Summary Measure | |
| | | 8.1.3. Population of Interest | |
| | | 8.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 8.1.5. Statistical Analyses / Methods | |
| ۵ | ΜΔΤΕΙ | RNAL AND INFANT ANALYSES | 22 |

| | 9.1. | Maternal Outcomes | |
|---|---|---|---|
| | | 9.1.1. Endpoints/Variables | |
| | | 9.1.2. Summary Measure | |
| | | 9.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 9.1.5. Statistical Analyses/ Methods | |
| | 9.2. | Infant Outcomes | |
| | J.Z. | 9.2.1. Endpoints/Variables | |
| | | 9.2.2. Summary Measure | |
| | | 9.2.3. Population of Interest | |
| | | 9.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 9.2.5. Statistical Analyses/ Methods | |
| 10 | VIROI | LOGY ANALYSIS | 25 |
| 10. | 10.1. | | |
| | 10.1. | I control of the cont | |
| | 10.2. | Statistical Analyses/Methods | |
| | 10.0. | Citationion / maryodo/motificati | |
| 11. | APPE | NDICES | 26 |
| | 11.1. | | |
| | | 11.1.1. Protocol Defined Schedule of Events | |
| | 11.2. | | |
| | | 11.2.1. Definitions of Assessment Windows for Analyses | |
| | | 11.2.2. Definitions of Assessment Windows for Inclusion in the PK | |
| | | Analysis | |
| | | 11.2.3. Stages of Pregnancy used for Pharmacokinetics | |
| | 44.0 | 11.2.4. Analysis visits in relation to pregnancy | 30 |
| | 11.3. | Appendix 3: Study Phases and Treatment Emergent Adverse | 0.4 |
| | | Events | |
| | | 11.3.1. Study Phases | 31 |
| | | 11.3.1.1. Treatment States for Laboratory, HIV | |
| | | Associated Conditions, Vital Signs, and | 24 |
| | | Genotypic and Phenotypic Data | 31 |
| | | | 24 |
| | | Therapy Medications Data | ا ک |
| | | 11.3.2. Treatment Emergent Flag for Adverse Events | |
| | 11.4. | Appendix 4: Data Display Standards & Handling Conventions | |
| | 11.4. | 11.4.1. Reporting Process | |
| | | 11.4.2. Reporting Standards | |
| | | 11.4.3. Reporting Standards for Pharmacokinetic | |
| | 11.5. | Appendix 5: Derived and Transformed Data | |
| | 11.0. | 11.5.1. General | |
| | | 11.5.2. Study Population | |
| | | 11.5.3. Efficacy | |
| | | 11.5.4. Safety | |
| | | 11.5.5. Pharmacokinetic | |
| | 11.6. | Appendix 6: Reporting Standards for Missing Data | |
| | | 11.6.1. Premature Withdrawals | |
| | | 11.6.2. Handling of Missing Data | |
| | | 11.6.2.1. Handling of Missing and Partial Dates | |
| | 11.7. | Appendix 7: Values of Potential Clinical Importance | |
| | | The second secon | |

# 2021N493381\_00 ING200336

### CONFIDENTIAL

| | 11.7.1. | Laboratory Values | 41 |
|--------|-----------------|-------------------------------------------|----|
| | 11.7.2. | Vital Signs | 41 |
| 11.8. | <b>Appendix</b> | c 8: Abbreviations & Trademarks | 42 |
| | | Abbreviations | |
| | 11.8.2. | Trademarks | 43 |
| 11.9. | Appendix | (9: Final (End of Study) Analysis | 44 |
| 11.10. | Appendix | c 10: List of Data Displays | 45 |
| | | Data Display Numbering | |
| | 11.10.2. | Mock Example Shell Referencing | 45 |
| | 11.10.3. | Deliverables | 45 |
| | 11.10.4. | Study Population Tables | 46 |
| | | Efficacy Tables | |
| | | Safety Tables | |
| | | Pharmacokinetic Tables | |
| | 11.10.8. | Pharmacokinetic Figures | 53 |
| | 11.10.9. | Virology Tables | 53 |
| | | .Maternal and Infant Assessment Tables | |
| | 11.10.11. | .ICH Listings | 55 |
| | | Non-ICH Listings | |
| 11.11. | | 11: Example Mock Shells for Data Displays | |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol: 200336

| Revision Chronology for Protocol: | | |
|---|---|---|
| GlaxoSmithKline | Date | Version |
| <b>Document Number</b> | | |
| 2013N166290 00 | 18-DEC-2013 | Original |
| 2013N166290 01 | 15-APR-2014 | Amendment No.: 01 |
| 2013N166290 02 | 23-APR-2014 | Amendment No.: 02 |
| 2013N166290 03 | 19-JUN-2018 | Amendment No.: 03 |
| Revision Chronology for RAP: | | |
| GSK2619619 ING200336<br>Reporting and Analysis Plan<br>(RAP) | 03-MAR-2021 | Original |
| GSK2619619 ING200336<br>Reporting and Analysis Plan<br>(RAP) Amendment 1 | 04-OCT-2021 | Amendment No.: 01 |

The main changes included in RAP amendment 01 are:

Tables for summary of absolute values for baseline and post-baseline of CD4+, Hematology and Chemistry are added at both Week 48 and End of Study analysis. Please see Appendix 10 for details.

Appendix 9 was added to describe the analysis that will be performed for the final end of study reporting.

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Pharmacokinetic Analysis: Log-transformed PK parameters except tmax will be analysed by analysis of variance | No ANOVA will be done. | Very few subjects<br>will be recruited |
| <ul> <li>Efficacy Endpoints for Infants:</li> <li>Proportion of subjects with plasma HIV-1 RNA &lt; 50 c/mL and &lt;400 c/mL over time.</li> <li>Absolute values and changes from Baseline in CD4+ T cell counts over time.</li> <li>Incidence of disease progression (HIV-associated conditions, acquired immunodeficiency syndrome [AIDS] and death).</li> </ul> | These data were not collected for Infants. | Inconsistencies within the protocol. The data for these endpoints were not collected in infants. |

# 2.2. Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| M | other |
| To describe the total plasma DTG PK parameters with the DTG/ABC/3TC FDC during Weeks 18-26, Weeks 30 – 36 of the third trimester of the pregnancy and 8-12 weeks postpartum | <ul> <li>Area under the concentration-time curve<br/>during a 24-hour interval at steady state<br/>[AUC24], maximal drug concentration<br/>[Cmax], drug concentration at the end of<br/>dosing interval [Cτ], Tmax, C0,<br/>apparent clearance [CL/F[, steady state<br/>volume of distribution [Vss/F] and the<br/>half-life [t½]) of DTG</li> </ul> |
| To further characterize the safety and<br>tolerability of DTG/ABC/3TC FDC<br>when used during pregnancy | <ul> <li>Incidence and severity of AEs and laboratory abnormalities.</li> <li>Absolute values and changes over time in laboratory parameters;</li> <li>Proportion of subjects who discontinue treatment due to AEs;</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Secondary Objectives | Secondary Endpoints |
| M | other |
| To assess the antiviral activity of the<br>DTG/ABC/3TC FDC when<br>administered during pregnancy | <ul> <li>Absolute values and change from<br/>Baseline HIV1 RNA over time.</li> <li>Proportion of subjects with plasma HIV-<br/>1 RNA &lt;50 and &lt;400 c/mL over time</li> </ul> |
| <ul> <li>To assess the immunologic activity of<br/>DTG/ABC/3TC FDC</li> </ul> | <ul> <li>Absolute values and change from<br/>Baseline in CD4+ cell count over time.</li> </ul> |
| Incidence of disease progression | <ul> <li>HIV-associated conditions, acquired<br/>immunodeficiency syndrome [AIDS]<br/>and death</li> </ul> |
| To assess the incidence of treatment –<br>emergent genotypic and phenotypic<br>resistance in subjects who meet<br>virologic withdrawal criteria | Treatment-emergent genotypic and<br>phenotypic resistance in subjects who<br>meet confirmed virologic withdrawal<br>criteria |
| To evaluate the unbound DTG concentrations in plasma during Weeks 18-26 and Weeks 30-36 of the pregnancy and 8-12 weeks postpartum | Unbound concentrations and Unbound<br>fraction at 3 and 24 hours post dose in<br>the third trimester and postpartum. |
| <ul> <li>To compare the DTG concentrations<br/>in plasma from cord blood with those<br/>in maternal plasma at the time of<br/>delivery</li> </ul> | <ul> <li>Total DTG concentrations in plasma<br/>from cord blood and those in maternal<br/>plasma at the time of delivery.</li> </ul> |
| To characterize pregnancy (maternal) outcomes | Pregnancy outcomes; Pregnancy risks |
| To characterize birth outcomes | <ul> <li>Birth outcomes (per pregnancy outcomes endpoint above)</li> </ul> |
| Infa | |
| To characterize infant outcomes at birth | Infant outcomes at birth |
| To characterize the safety of<br>DTG/ABC/3TC FDC to the<br>developing fetus | Proportion of pregnancies with and<br>without demonstrated congenital<br>malformations |

# 2.2.1. Study Design

| Overview of Study Design and Key Features | |
|---|---|
| Design<br>Features | <ul> <li>This is a single arm open-label interventional study for women who<br/>become pregnant while participating in ING117172 on the<br/>DTG/ABC/3TC FDC treatment arm.</li> </ul> |
| Dosing | <ul> <li>All subjects will be administered DTG 50 mg/ABC 600 mg/3TC 300<br/>mg FDC tablet administered once daily.</li> </ul> |
| Time & Events | Refer to Appendix 1: Schedule of Activities |

| Overview of S | Overview of Study Design and Key Features |
|---|---|
| Treatment<br>Assignment | <ul> <li>Subjects will initiate therapy with DTG/ABC/3TC FDC following<br/>confirmation of fulfilment of study entry criteria. A unique treatment<br/>number will be assigned for each subject participating in the study.<br/>Subjects who are enrolled into the trial and subsequently withdrawn<br/>may not be re-screened.</li> </ul> |
| Interim<br>Analysis | <ul> <li>No interim analysis was planned, however protocol allowed further<br/>data cuts and analyses to be conducted as necessary to support<br/>regulatory requests, submissions and/or publications. The study<br/>recruitment was terminated early which triggered reporting of the<br/>primary endpoint.</li> </ul> |

# 2.3. Statistical Hypotheses / Statistical Analyses

This is a single arm open-label interventional study for women who become pregnant while participating in ING117172. No formal hypotheses testing will be performed.

## 2.4. Interim Analyses

No interim analyses were formally planned, however the protocol allows further data cuts and analyses are conducted as necessary to support regulatory requests, submissions and/or publications. The planned analyses will be performed after the completion of the following sequential steps:

- 1. Subjects are considered to have completed the study after completing the postpartum evaluation approximately 8-12 weeks post-delivery. The primary outcome analyses will take place after the last subject enrolled gives birth and completes their last visit.
- 2. All required database cleaning activities have been completed.

# 2.5. Final Analyses

Subjects may continue to receive DTG/ABC/3TC FDC after completion of the primary endpoint assessments, until study medications are locally approved and commercially available (or they meet a criteria for withdrawal). During this time, subjects will be monitored every 12 weeks to ensure they continue to derive clinical benefit from DTG/ABC/3TC FDC.

A final End-of-Study analysis will be conducted when all subjects have completed the study and final database release (DBR), source data lock (SDL) and database freeze (DBF) have been declared by Data Management.

# 3. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All subjects<br>Screened | All participants who were screened for eligibility | Study Population |
| Enrolled | All participants who passed screening and entered the study | Study Population |
| Safety/ITT-E | All participants who received at least one dose of study treatment. | <ul><li>Study Population</li><li>Safety</li><li>Efficacy</li></ul> |
| Pharmacokinetic<br>(PK) | <ul> <li>All participants in the Safety population who had at least<br/>1 non-missing PK assessment (Non-quantifiable [NQ]<br/>values will be considered as missing values)</li> </ul> | • PK |
| | Note: PK samples that may be affected by protocol<br>deviations will be reviewed by the study team to<br>determine whether or not the sample will be excluded. | |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

## 3.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) and non-important COVID-19 related protocol deviations will be listed.

# 4. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 4.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | Data Displays for Reporting | | |
| Code | Code Description Description Order | | |
| Α | DTG/ABC/3TC FDC once daily | DTG/ABC/3TC | 1 |

No subgroup analysis will be done.

#### 4.2. Baseline Definitions

For all endpoints (unless otherwise stated) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data are missing no derivation will be performed and baseline will be set to missing.

Unless otherwise specified, the baseline definitions specified in the table below will be used for derivations for endpoints/parameters and indicated on listings.

| Definition | Reporting Details |
|------------------------|-----------------------------------------------------|
| Change from Baseline | Post-Dose Visit Value Baseline |
| % Change from Baseline | 100 x [(Post-Dose Visit Value Baseline) / Baseline] |

#### 4.3. Multicentre Studies

There are no planned adjustments made for multiple centres in this study.

## 4.4. Examination of Covariates, Other Strata and Subgroups

No covariates, Strata or Subgroups will be considered for descriptive summaries or Statistical analysis.

# 4.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

# 2021N493381\_00 ING200336

### CONFIDENTIAL

| Section | Component |
|---------|----------------------------------------------------------------|
| 11.2 | Appendix 2 : Assessment Windows |
| 11.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Reporting Standards for Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |

# 5. STUDY POPULATION ANALYSES

# 5.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Enrolled and ITT-E population.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 9: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data Display's Generated | |
|---|---|---|
| | Table | Listing |
| Randomisation | | • |
| Randomisation | | Y |
| Subject Disposition | | |
| Study Populations | | Y |
| Subject Recruitment by country and site ID | Υ | Y |
| Disposition (overall and by relationship to COVID-19 Pandemic) | Υ | |
| Reasons for Withdrawal | | Y |
| Study Visit Dates | | Y |
| Protocol Deviations | | |
| Important Protocol Deviations | | Y |
| Non-Important COVID-19 related Protocol Deviations | | Υ |
| <b>Demography and Baseline Characteristics</b> | | |
| Demographic Characteristics | Υ | Y |
| Age Ranges | Υ | |
| Race | Υ | Y |
| CDC Classification of HIV infection at Baseline | | Υ |
| Cardiovascular Risk Assessments at Baseline | | Υ |
| History of Cardiac Therapeutic Procedures | | Υ |
| Cardiovascular Events at Baseline | | Υ |
| Maternal History (Pregnancy History) | | Y |
| Medical Conditions, Concomitant Medications & Ant | iretroviral Therapy | |
| Medical Conditions (Current and Past) | | Y |
| Concomitant Medications (non-ART) | | <b>Y</b> [1] |
| Prior and Concomitant ART Medications | | Y [2] |

| Display Type | Data Display's Generated | |
|-------------------------|--------------------------|---------|
| | Table | Listing |
| Other | | |
| Investigational Product | | Y |

#### **Notes:**

- Y = Display Generated
- 1. One listing for concomitant non-ART medications and one listing showing the relationship between verbatim text, ingredient and ATC Level 1.
- 2. One listing for Prior ART, one listing for concomitant ART and one listing showing the relationship between verbatim text, ingredient, combination and ATC Level 4.

## 6. EFFICACY ANALYSES

## 6.1. Endpoint / Variables

#### Mother

- Absolute value and change from baseline in HIV-1 RNA over time
- Proportion of subjects with plasma HIV-1 RNA <50 and <400 c/mL over time
- Absolute value and change from baseline in CD4+ Cell count over time
- Disease progression and HIV associated conditions

## 6.2. Summary Measure

Efficacy data will be presented in tabular form and will be summarized descriptively by visit.

## 6.3. Population of Interest

The efficacy analyses will be based on the Intent-To-Treat- Exposed population, unless otherwise specified.

## 6.4. Strategy for Intercurrent (Post-Randomization) Events

Not applicable.

# 6.5. Efficacy Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 6.1 will be listed and summarised.

Table 3 Overview of Planned Efficacy Analyses

| Endpoints | Absolute | | | Change from Baseline | | | ine | |
|---|---|---|---|---|---|---|---|---|
| | Sumr | Summary | | idual | Summary | | Individual | |
| | T | F | F | L | Т | F | F | L |
| Quantitative Plasma H | IIV-1 RNA | | | | | | | |
| Observed over time | | | | Υ | Y | | | |
| Proportion of<br>Subjects with Plasma<br>HIV-1 RNA <400<br>copies/mL | Y | | | | | | | |
| Proportion of<br>Subjects with Plasma | Y | | | | | | | |

| Endpoints | Absolute | | | Change from Baseline | | | ine | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Summary Individual | | Summary | | Individual | |
| | T | F | F | L | Т | F | F | L |
| HIV-1 RNA <50<br>copies/mL | | | | | | | | |
| CD4+ Cell Count | | | | | | | | |
| Observed over time | Y | | | Υ | Y | | | |
| Post-baseline HIV-1 Disc | ease Progr | ession | | | | | | |
| Incidence of disease progression <sup>[1]</sup> | Y | | | | | | | |

**NOTES:** L = Listing, Y = Yes display generated.

<sup>1.</sup> HIV-associated conditions, acquired immunodeficiency syndrome [AIDS] and death

# 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

# 7.1. Adverse Events Analyses

The details of the planned displays are provided in Appendix 9: List of Data Displays.

Table 4 Overview of Planned Safety Analyses

| | A | bsolute |
|---|---|---|
| Display Type | Summary | Individual |
| | T | L |
| Exposure Data | | Y |
| All Adverse Events | | Y |
| Non-Fatal serious Adverse<br>Events | | Y |
| Non-Serious Drug-Related<br>Adverse Events by Overall<br>Frequency | Y | |
| All Adverse Events by System<br>Organ Class, Preferred Term and<br>Maximum Toxicity | Y | |
| Non-serious Adverse Events by<br>System Organ Class and<br>Preferred Term (Number of<br>Subjects and Occurrences) | Y | |
| Grade 2-4 Adverse Events by<br>Overall Frequency | Y | |
| Serious Adverse Events by<br>System Organ Class and<br>Preferred Term (Number of<br>Subjects and Occurrences) | Y | |
| Serious Fatal and Non-Fatal<br>Drug-Related Adverse Events by<br>Overall Frequency | Y | |

| | Absolute | |
|---|---|---|
| Display Type | Summary | Individual |
| | T | L |
| Reasons for Considering as a<br>Serious Adverse Event | | Y |
| Adverse Events Leading to<br>Permanent Discontinuation of<br>Study Treatment or Withdrawal<br>from Study | Y | Y |
| Relationship of Adverse Event<br>System Organ Classes, Preferred<br>Terms, and Verbatim Text | | Y |
| COVID-19 Assessments and Symptom assessments | | Y |

**NOTES:** • T = Table, L = Listing, Y = Yes display generated.

# 7.2. Clinical Laboratory and Other Safety Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests and Urinalysis, and non-laboratory safety test results including vital signs, cardiovascular events and suicidality monitoring tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 9: List of Data Displays.

| Endpoint | | Absolute | | С | Change from Baseline | | | | Max Post BL | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | Summary | | Summary Individual | | Stats Analysis | | Summary | | Summary | | |
| | T | F | F | L | T | F | L | T | F | T | F | L |
| Laboratory values | | | | | | | | | | | | |
| Clinical Chemistry | | | | Υ | | | | Y | | Υ | | |
| Haematology | | | | Υ | | | | Y | | Υ | | |
| Urinalysis | | | | Υ | | | | Y | | | | |
| Non-Laboratory va | lues | | | | | | | | | | | |
| Vital Signs | | | | Y | | | | | | | | |
| Suicidal Ideation | | | | Υ | | | | | | | | |
| and Behaviour | | | | | | | | | | | | |
| Data | | | | | | | | | | | | |
| Others | | | | | | | | | | | | |
| COVID-19 | | | | Υ | | | | | | | | |
| Symptom and | | | | | | | | | | | | |
| assessments | | | | | | | | | | | | |

**NOTES**: T=Table, F=Figure, L = Listing, Y = Yes display generated

#### 8. PHARMACOKINETIC ANALYSES

## 8.1. Primary and Secondary Pharmacokinetic Analyses

### 8.1.1. Endpoint / Variables

Pharmacokinetic parameters will be determined from the plasma concentration-time data, as data permits.

#### **Primary PK Analysis Endpoints:**

DTG AUC(0- $\tau$ ), Cmax, C $\tau$ , CL/F, Vss/F, and  $t_2$  based on intensive PK sampling during the second and third trimesters of pregnancy (Weeks 18-26 and 30-36) and at 8-12 weeks postpartum will be determined, as data permits.

#### **Secondary PK Analysis Endpoints**

- C0 and Tmax based on intensive PK sampling during the second and third trimesters of pregnancy (Weeks 18-26 and 30-36) and at 8-12 weeks postpartum
- C3h,u and C24h,u and fu at the PK visits during the second and third trimesters and at 8-12 weeks postpartum
- Total DTG concentrations in plasma from cord blood compared to those in maternal plasma at the time of delivery.

## 8.1.1.1. Drug Concentration Measures

All PK concentration summary and listing displays will be based on Pharmacokinetic population. Concentrations of DTG in plasma will be listed and summarized according to GSK standards, where applicable (Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Standards for Pharmacokinetic).

DTG concentration listings for the PK population will be sorted by subject and time relative to dose, noting the study visit; summaries will be presented by time relative to dose at each PK visit -Weeks 18-26 and Weeks 30-36 of pregnancy, and at 8-12 weeks post-partum (See Appendix 2: Section 11.2.3 for details). At each PK visit, samples will be collected prior to dosing and at 1,2, 3, 4, 6, 8, 12 and 24 hours post dosing. The predose sample should be collected within 15 minutes prior to the dose on the day of PK visit. DTG concentrations in plasma from cord blood will also be collected at the time of delivery will be compared with those in maternal plasma at the time of delivery.

#### 8.1.1.2. Derived Pharmacokinetic Parameters

PK analysis will be the responsibility of the Clinical PK Modeling & Simulation department within GlaxoSmithKline. Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 5.2 or higher. All calculations of non-

compartmental parameters will be based on actual sampling times recorded during the study. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

Table 5 Table of Derived PK Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | DTG Area under the plasma concentration time curve at steady state during a dosing interval |
| C0 | DTG Pre-dose plasma concentration |
| Cmax | DTG maximum observed plasma concentration determined directly from the concentration-time data. |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Сτ | Drug concentration at the end of dosing interval. |
| CL/F | Apparent oral clearance. |
| Vss/F | Apparent volume of distribution after extravascular (e.g., oral) administration. |
| t½ | DTG half-life. |
| C3h,u | Unbound DTG concentration in plasma at 3 hours post dose |
| C24h, u | Unbound DTG concentration in plasma 24 hours post dose |
| Weight Normalised<br>CL/F | Apparent oral clearance |
| Weight Normalised<br>Vss/F | Apparent volume of distribution after extravascular (e.g., oral) administration |
| fu3h and fu24h | Unbound fraction at 3 hours and 24 hours post dose, calculated as: |
| | fu Cunbound/Ctotal |
| | where Cunbound and Ctotal are the unbound and total concentration of DTG in plasma, respectively. |

## 8.1.2. Summary Measure

Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively by time relative to dose at each PK visit -Weeks 18-26 and Weeks 30-36 of pregnancy, and at 8-12 weeks post-partum (See Appendix 2: Section 11.2.3 for details).

## 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

#### 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

Not Applicable.

## 8.1.5. Statistical Analyses / Methods

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

Table 6 provides an overview of the planned analyses, with full details being presented in Appendix 9: List of Data Displays.

Table 6 Overview of Planned Pharmacokinetic Analyses

| | | Untrar | sforme | i | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| <b>End Point</b> | Summary | | Indiv | vidual | Sum | mary | Individual | |
| | T | F | F | L | T | F | F | L |
| PK Concentrati | PK Concentrations | | | | | | | |
| Plasma DTG<br>Concentrations | Y | Y | Y | Y | Y | Y | Y | |
| PK Parameters | | | | | | | | |
| Plasma DTG<br>Parameters | Y | | | Y | Y | | | |

Note: T Table, F Figure, L Listing, Y = Yes display generated

## 9. MATERNAL AND INFANT ANALYSES

#### 9.1. Maternal Outcomes

## 9.1.1. Endpoints/Variables

- Pregnancy outcomes variables: Spontaneous loss/miscarriage, Elective termination, Still birth, Live birth. In case of Live birth applicable Birth outcome categories will be listed.
- Maternal History
- Previous and Current Pregnancy risk assessment

## 9.1.2. Summary Measure

Current Maternal data will be summarised over each maternal outcome.

#### 9.1.3. Population of Interest

The Maternal Outcome analysis will be based on the Safety population, unless otherwise specified.

#### 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

Not applicable.

## 9.1.5. Statistical Analyses/ Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, all endpoints / variables defined in Section 9.1.1 will be listed. The pregnancy outcomes will be summarised.

#### 9.2. Infant Outcomes

#### 9.2.1. Endpoints/Variables

Infant outcome variables:

- Infant gestational age,
- Gestational length,
- Gestational weight (including percentiles, SGA, AGA, LGA, IUGR [IUGR in case of SGA only])
- Head circumference
- APGAR (Appearance, Pulse Rate, Grimace Reflex, Activity, Respiration) one and five minute scores
- Presence or absence of major congenital abnormalities at birth.
- HIV Status of Infant at 8-12 week postpartum visit

## 9.2.2. Summary Measure

The Infant data will be summarised over each outcome.

### 9.2.3. Population of Interest

The Infant Outcome analysis will be based on the Safety Population, unless otherwise specified.

### 9.2.4. Strategy for Intercurrent (Post-Randomization) Events

Not applicable.

## 9.2.5. Statistical Analyses/ Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.2.1 will be listed and summarised.

## 10. VIROLOGY ANALYSIS

## 10.1. Endpoints/Variables

Treatment-emergent genotypic and phenotypic resistance in subjects who meet confirmed virologic withdrawal criteria

## 10.2. Population of Interest

The virology analyses will be based on the ITT-E population, unless otherwise specified.

# 10.3. Statistical Analyses/Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoint defined in Section 10.1 will be summarised.

# 11. APPENDICES

# 11.1. Appendix 1: Schedule of Activities

# 11.1.1. Protocol Defined Schedule of Events

| Procedures | Screen'." | Day 1 | Ante partum | Delivery | Post-Partum | Continuation<br>Phase | Withdrawal | Follow-up <sup>12</sup> |
|---|---|---|---|---|---|---|---|---|
| | | | Monthly – every 4<br>weeks | | 8-12 weeks<br>post delivery | Every 12 weeks<br>after Post<br>Partum Visit | | |
| Written Informed Consent | X | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | X | | | | | | |
| Subject Demography | X | | | | | | | |
| Medical History <sup>1</sup> | | X | | | X | X | | |
| Concurrent medical conditions | | X | | | | | | |
| CDC HIV-1 classification | | X | | | | | | |
| HIV-associated conditions | | | X | Х | X | X | X | X |
| Cardiovascular risk<br>assessment <sup>2</sup> | * | | | | | | | |
| Prior Art history | * | | | | | | | |
| Gravidity Maternal history | | X | | | | | | |
| Pregnancy risk assessment | X | X | X | | | | | |
| Uteroplacental Outcomes<br>at Delivery <sup>a</sup> | | | | Х | | | | |
| Infant Outcomes4 | | | | X | X | X | | X |
| Concomitant Medication | X | Х | X | Х | X | X | X | X |
| Limited Physical<br>Examination <sup>6</sup> | | X | X | | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X |

| Procedures | Screen'." | Day 1 | Ante partum | Delivery | Post-Partum | Continuation<br>Phase | Withdrawal | Follow-up <sup>12</sup> |
|---|---|---|---|---|---|---|---|---|
| | | | Monthly – every 4<br>weeks | | 8-12 weeks<br>post delivery | Every 12 weeks<br>after Post<br>Partum Visit | | |
| Serious Adverse Events® | X | X | X | <b>X</b> 6 | Х | X | X | X |
| Pharmacokinetic<br>Sampling <sup>7</sup> | | | Χε | X | X | | | |
| Cord & maternal blood<br>sample <sup>8</sup> | | | | X | | | | |
| Columbia Suicidality<br>Severity Rating Scale | | X | X | | X | X | Х | |
| Laboratory Assessments | | | | | | | | |
| Pregnancy Assessment | | X | | | Х | X | | |
| Hematology | ** | ** | X | | Х | Х | X | X |
| Clinical Chemistry | ** | ** | X | | X | X | X | X |
| Urinalysis. Including | ** | | X | | X | X | | X |
| dipstick for protein<br>analysis | | | | | | | | |
| Quantitative plasma HIV-1<br>RNA <sup>10</sup> | ** | ** | X | X | X | X | X | |
| Lymphocyte subsets | ** | ** | X | <b>X</b> 6 | X | X | | X |
| PGx Sampling <sup>11</sup> | | X | | | | | | |
| Plasma for storage12 | X | X | X | X | X | X | X | X |
| Dispense IP | | X | X | X | X | Х11 | | |

<sup>\*</sup>Baseline information, including cardiovascular risk and prior ART therapy will be transferred from ING117172 to serve as baseline/screening data in this study.

Gravidity: Maternal history and pregnancy risk assessment may occur at either Screening or Day 1 visit.

1. Medical History includes any changes in smoking status

inING200336.

- 2. Assessment for cardiovascular risk will include height, weight, blood pressure, smoking history, medical conditions and will have previously been collected in ING117172
- 3. Assessment of pregnancy outcomes (e.g., spontaneous losses, induced abortions, still births, pre-term births, preeclampsia)
- 4. Assessment of maternal and infant outcomes, including live births, gestational age, presence or absence of major congenital abnormalities, and infant height, weight, [including percentiles, SGA, AGA, LGA, IUGR], head circumference, and presence or absence of major congenital abnormalities at birth. If known, HIV status of the infant will be collected at the 8-12 week post-partum visit.
- 5. Limited physical examination to include blood pressure at Baseline (recorded in eCRF), heart rate and weight at each visit (recorded in eCRF at Baseline and on lab requisition at all visits) for determination of CrCL. Blood pressure to be measured after resting in a semi-supine position for at least 5 minutes.
- 6. From the time a subject consents to participate in ING200336 and administration of IP at Day 1, only SAEs assessed as related to study participation (e.g., study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication, will be recorded in the eCRF for ING200336. Only SAEs related to study participation or to a concomitantly administered GSK or ViiV product will be collected between obtaining informed consent and administration of IP at Day 1.
  Note: At the time of the Withdrawal visit in ING117172 if there is an ongoing, unresolved adverse event (AE) and/or serious adverse event (SAE) it will be left in ING117172 as unresolved and transcribed as medical history in ING200336. If the AE and/or SAE worsen after enrollment into ING200336 it will be recorded on the AE/SAE forms
- 7. Intensive PK visit: The PK evaluations should be scheduled for study visits at Weeks 18-26, Weeks 30-36 and 8-12 weeks postpartum. The DTG dose on serial PK sampling days is to be given with a light meal/snack PK should be

<sup>\*\*</sup>HIV-1 RNA, lymphocyte subset, and laboratory assessment (hematology, chemistry, and urinalysis including a dipstick) data collected at the ING117172 unscheduled or last visit within 28 days of learning of the pregnancy will be transferred to serve as screening data in this study. The ING117172 Withdrawal visit will serve as the ING200336 Day 1.

- scheduled so that witnessed dosing of DTG/ABC/3TC FDC is as close as possible to 24 hours (generally 22-26 hours) after the previous dosing. The PK visit should be re-scheduled if the subject took their morning dose prior to coming into the clinic on the PK sampling day. See SPM for additional details.
- 8. If feasible, a cord and maternal blood sample will also be collected at delivery and if possible within 30 minutes of each other.
- 9. Suicidality Questionnaire will be conducted q 12 weeks during the Continuation Phase.
- 10. HIV-1 RNA and lymphocyte to be drawn within 24 hours of delivery and on the day of the post-partum PK evaluation.
- 11. The PGx sample should be collected at Day 1 if not collected during participation in ING117172, however this sample may be collected at any time during the study.
- 12. Plasma samples for storage will be collected at each visit for possible future analyses (including but not limited to HIV-1 RNA genotypic and phenotypic analyses in confirmed cases of subject withdrawal, HIV-1 RNA levels, when samples are lost or arrive at the laboratory unevaluable, and immunological parameters.)
- 13. Only for subjects who continue DTG/ABC/3TC and are seen in the clinic every 12 weeks until DTG/ABC/3TC is commercially available locally. Note: after delivery, subjects must use one of the contraception methods to avoid a 'new' pregnancy
- 14. A Follow up visit may be conducted approximately 4 weeks after the last dose of study provided IP, and is required only if the subject has ongoing SAEs or non-serious AEs (as outlined in the SPM) at the last on study visit. The assessments performed should reflect what is considered medically necessary to assess the event(s).

## 11.2. Appendix 2: Assessment Windows

Laboratory data and vital signs will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

A window around a target Study Day will typically include all days from the midpoints between it and the target Study Days of the previous and the proceeding visits. In general, the nominal target study day for week w is (7\*w)+1.

## 11.2.1. Definitions of Assessment Windows for Analyses

| Analysis Set | Parameter | Target | Analysis | Window | Analysis |
|---|---|---|---|---|---|
| / Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| All | All | | | | Screening |
| | | 1 | | | Day 1 |
| | | 29 | 2 | 42 | Week 4 |
| | | 57 | 43 | 70 | Week 8 |
| | | 85 | 71 | 98 | Week 12 |
| | | 113 | 99 | 126 | Week 16 |
| | | 141 | 127 | 154 | Week 20 |
| | | 169 | 155 | 182 | Week 24 |
| | | 197 | 183 | 210 | Week 28 |
| | | 225 | 211 | 238 | Week 32 |
| | | 253 | 239 | 266 | Week 36 |
| | | 281 | 267 | 294 | Week 40 |
| | | 337 | 295 | 378 | Week 48 |
| | | 7*w+1 | 7*w-41 | 7*w+42 | Week w,<br>w=52, 64,<br>76, |
| | | Study Day of last dose<br>+ 28 | >Study Day<br>of last dose<br>+1 | >Study Day<br>of last dose<br>+1 | Follow-up |

#### **NOTES:**

- For parameters which are not scheduled to be assessed at particular visits, the all-inclusive windows defined will still be used.
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings.

# 11.2.2. Definitions of Assessment Windows for Inclusion in the PK Analysis

The windows for inclusion of PK samples in summary statistics for all PK visits will be as follows:

- Samples collected 15 minutes prior to dose for pre-dose sample
- O Samples collected within  $\pm 15$  min of the 1h and 2h time points
- O Samples collected within  $\pm$  30 min of the 3h, 4h, 6h time points
- O Samples collected within  $\pm$  1h for the 8h and 12h time points
- O Samples collected within  $\pm$  2h for the 24 h time point

### 11.2.3. Stages of Pregnancy used for Pharmacokinetics

| Stage | Weeks | |
|-------------|-------------|-------|
| Ante-Partum | Trimester 2 | 18-26 |
| | Trimester 3 | 30-36 |
| | Delivery | |
| | Post-Partum | |

#### NOTES:

- Delivery is a single day.
- Post-partum PK assessment is done 8-12 weeks after delivery

## 11.2.4. Analysis visits in relation to pregnancy

In addition, an analysis visit in relation to pregnancy is derived, which will also be listed in the listings.

- For the screening, delivery and post-partum visits, the same scheduled visit is used.
- For the Day 1 and ante-partum visits, the corresponding gestation weeks from reproductive system findings is used.
- For the subsequent post-partum visits, the analysis visit in relation to pregnancy is derived by (visit day of subsequent post-partum visit visit day at post-partum)/7.

# 11.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

## 11.3.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to Study Visits.

# 11.3.1.1. Treatment States for Laboratory, HIV Associated Conditions, Vital Signs, and Genotypic and Phenotypic Data

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date + 1 |

#### 11.3.1.2. Treatment States for Prior/Concomitant/Post-Therapy Medications Data

- Prior medications are those taken (i.e., started) before the start date of investigational product.
- Concomitant medications are those taken (i.e., started or continued) at any time between the start date and stop date of IP, inclusive. Prior medications that were continued during this period are also considered as concomitant medications.
- Post-treatment medications are those started after the stop date of IP.
   Concomitant medications that were continued during this period are also considered as post-treatment medications.

It will be assumed that medication has been taken on the date in which it is reported as started or stopped. Also, for any medication starting on the same date as IP, it will be assumed that the medication was taken after the subject started taking IP.

ART medications will also be classified as prior, concomitant and/or post-treatment according with the following modifications:

- ART starting on study treatment stop date will be considered as only posttreatment and not concomitant. It is expected that after discontinuation of study treatment, a subject may immediately begin taking another ART.
- ART stopping on study treatment start date will only be considered as prior and not concomitant.
- Any ART entered on the Prior ART eCRF with partial end date will be assumed to have finished before Screening.

| | | re-<br>tment | | On-t | reatment | | Pos | st-treatr | nent | Prior | Conco-<br>mitant | Post |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (a) | X | Х | | | | | | | | Υ | N | N |
| (b) | X | | | | X | | | | | Υ | Υ | N |
| (c) | X | | | | | | | | X | Υ | Υ | Υ |
| (d) | | | | х | X | | | | | N | Υ | N |
| (e) | | | پو ا | Х | | ø | Ŧ | | X | N | Υ | Υ |
| (f) | | | Dat | | | Dat | ate | X | X | N | N | Υ |
| (g) | ? | X | IP Start Date | | | IP Stop Date | IP Stop Date+1 | | | Υ | N | N |
| (h) | ? | | St | | X | St | Sto | | | Y* | Υ | N |
| (i) | ? | | _ ₽ | | | _ | Ы | | X | <b>Y</b> * | Y* | Υ |
| (j) | x | | | | | | | | ? | Υ | Υ** | Y** |
| (k) | | | | х | | | | | ? | N | Υ | Y** |
| (1) | | | | | | | | X | ? | N | N | Υ |
| (m) | ? | | | | | | | | ? | Y*** | Y*** | Y*** |
| (n) | X | | X | | | | | | | Υ | Υ | N |
| (o) | ? | | Х | | | | | | | Y* | Υ | N |
| (p) | | | Х | | X | | | | | N | Υ | N |
| (q) | | | Х | | | Х | | | | N | Υ | N |
| (r) | | | | | | Х | | | X | N | Υ | Υ |
| (s) | | | | | | X | | | ? | N | Υ | Y** |
| (t) | | | | | | | X | | X | N | N | Υ |
| (u) | | | | | | | X | | ? | N | N | Υ |
| (v) | | | | Х | | | X | | | N | Υ | Υ |

x = start/stop date of medication

#### 11.3.1.3. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date |
| Onset Time Since<br>1st Dose (Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 |

<sup>? =</sup> missing start/stop date of medication

<sup>\*</sup> If a medication is stopped On-treatment or Post-treatment and no start date is recorded it will be assumed that the medication was ongoing from the Pre-treatment phase

<sup>\*\*</sup> If a medication is started Pre-treatment or On-treatment and no stop date is recorded then usage will be assumed to be ongoing for the remainder of the study

<sup>\*\*\*</sup> If a medication has no start or stop date it will be assumed that the medication was ongoing from the Pre-treatment phase to the Post-treatment phase

| Treatment State | Definition |
|-----------------|-----------------------------------------|
| | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on CRF. |

#### NOTES:

- In the case of a completely missing start date, the event will be considered to have started On-treatment unless
  an end date for the AE is provided which is before start of investigational product; in such a case the AE is
  assigned as Pre-treatment.
- If the IP Stop Date is missing, then any event with a start date on or after IP Start Date will be considered to be On-treatment.
  - If the start date of the AE is after IP Stop Date but has been recorded as potentially related to IP, then it will be classified as On-treatment.

## 11.3.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Emergent | Emergent refers to AE Severity/ Lab toxicity that develops or increases in intensity after baseline |

#### NOTES:

- If the study treatment stop date is missing, then the AE/ Lab toxicity will be considered to be
  On-Treatment unless an end date for the AE/ Lab toxicity is provided which is before start of
  investigational product; in such a case the AE/ Lab toxicity is assigned as Pre-treatment.
- Time of study treatment dosing and start/stop time of AEs/ Lab toxicity should be considered, if collected.

# 11.4. Appendix 4: Data Display Standards & Handling Conventions

## 11.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Compound | :\ARPROD\GSK2619619\ING200336\Documents\final 01(SAC) |
| Analysis Datasets | |

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1 or above).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented as SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts.

## 11.4.2. Reporting Standards

#### General

 The current GSK Statistical Display Standards in the GSK Standards Library (IDSL) will be applied for reporting, unless otherwise stated (Library Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK Statistical Display Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the GSK Standard Statistical Display Principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to GSK Standard Statistical Display Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

| Unscheduled Visits | |
|---|---|
| Unscheduled visits will be included in listings. | |
| Unscheduled visits will be assigned to a study visit using the all-inclusive windows defined in Section | |
| 11.2.1 | |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to GSK Standard Statistical Display Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| <ul> <li>Refer to GSK Standard Statistical Display Principals 7.01 to 7.13.</li> </ul> | |

# 11.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to Standards for the Transfer and Reporting of PK Data document. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to the GSK Standard PK Display Standard. Refer to the GSK Standard Statistical Display Principle 6.06.1. Note: If any concentration value is not calculable because of NQs, it will be excluded (set to missing) from the PK concentration Summary tables and Graphical displays and show as NQ in Listings. Refer to VQD-GUI-000722 (6.0) (Non-Compartmental Analysis of Pharmacokinetic Data) for handling of values below the Quantification Limit. |
| Pharmacokinetic Parameter Derivation | |
| PK Parameter to be<br>Derived by<br>Programmer | The PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using WinNonLin v 5.2 or above. All calculations of non-compartmental parameters will be based on actual sampling times. |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | If any PK parameter is not calculable because of NQs, it will be excluded (set to missing) from the PK parameter summary. Refer to VQD-GUI-000722 (6.0) (Non-Compartmental Analysis of Pharmacokinetic Data) for handling of values below the Quantification Limit. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to GSK Standard PK Display Standard. |
| Untransformed PK parameter | tmax (TMAX), t1/2 |

## 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

#### Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 11.2.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from initial study treatment start date:
  - Ref Date = Missing 
    → Study Day = Missing
  - Ref Date < Treatment Start Date → Study Day = Ref Date -Treatment Start Date
  - Ref Data ≥ Treatment Start Date → Study Day = Ref Date (Treatment Start Date) +
  - Note that Treatment Start Date is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### **Post Baseline**

Post-baseline refers to the combined time periods of On-treatment and Post-treatment.
 Post-baseline may be further specified according to phase of the study: Antepartum,
 Delivery, Postpartum or Continuation.

## 11.5.2. Study Population

#### Extent of Exposure

- Number of days of exposure to study drug will be calculated based on the formula:
- Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:
- Cumulative Dose = Sum of (Number of Davs x Total Daily Dose)
- If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Since only year of birth is recorded for subjects (day and month are not recorded), for the purpose of calculating age, day and month of birth will be imputed as '30th June'.
### 11.5.3. Efficacy

#### **HIV-1 RNA**

Plasma for quantitative HIV-1 RNA will be collected. Methods to be used may include but are not limited to the Abbott RealTime HIV-1 Assay lower limit of detection (LLOD) 40 c/mL. In some cases (e.g., where the HIV-1 RNA is below the LLOD for a given assay) additional exploratory methods may be used to further characterize HIV-1 RNA levels.

#### Lymphocyte

#### CD4+ Cell Count

Absolute CD4+ lymphocyte counts will be collected for assessment by flow cytometry.

### 11.5.4. Safety

#### **Adverse Events**

#### AE Severity – DAIDS Grading.

- The DAIDS grading for severity of clinical adverse events will be performed.
- See protocol for DAIDS grading criteria.

### **Suicidality Monitoring**

 Treatment emergent assessment of suicidality will be monitored during this study using the Columbia Suicide-Severity Rating Scale.

#### **Laboratory Parameters**

#### Lab Toxicities – DAIDS Grading

- The DAIDS grading for severity of clinical adverse events will be performed.
- See protocol for DAIDS grading criteria

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has
  a non-detectable level reported in the database, where the numeric value is missing, but
  typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than
  x in the comment field) is present, the number of significant digits in the observed values will
  be used to determine how much to add or subtract in order to impute the corresponding
  numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</li>

# 11.5.5. Pharmacokinetic

# PK Parameters

- The PK Population will include all subjects who undergo PK sampling and have evaluable PK assay results.
- See Table 5 for derived Pharmacokinetic parameters

# 11.6. Appendix 6: Reporting Standards for Missing Data

# 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as: Subjects are considered to have completed the study after completing the postpartum evaluation.</li> <li>Withdrawn participants were not replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables, listings and figures, unless otherwise specified.</li> </ul> |

# 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

### 11.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in participant listing displays.</li> </ul> |
| Adverse<br>Events | <ul> <li>Imputations in the adverse events dataset are used for slotting events to the appropriate study time periods and for sorting in data listings.</li> <li>Partial dates for AE recorded in the CRF will be imputed using the following conventions:</li> </ul> |
| | If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month. Else if study treatment start date is not missing: |
| | <ul> <li>Missing start day and month</li> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> </ul> </li> </ul> |

| Element | Reporting Detail | |
|---|---|---|
| | Missing stop day Missing stop day | If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1. Else set start date = study treatment start date. Else set start date = January 1. Last day of the month will be used. No Imputation |
| | and month Completely missing start/end date | No imputation |
| | Completely miss | ing start or end dates will remain missing, with no imputation applied. |
| Concomitant<br>Medications/<br>Medical | | for any concomitant medications recorded in the CRF will be imputed lowing convention: |
| History | Missing start day | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing end day | A '28/29/30/31' will be used for the day (dependent on the month and year) |
| | Missing end day and month | A '31' will be used for the day and 'Dec' will be used for the month. |
| | Completely missing start/end date | No imputation |
| | The recorde | d partial date will be displayed in listings. |

# 11.7. Appendix 7: Values of Potential Clinical Importance

# 11.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Hematocrit | Ratio of | | | 0.54 |
| nematocht | 1 | $\Delta$ from BL | -0.075 | |
| Haamaglahin | g/L | | | 180 |
| Haemoglobin | | $\Delta$ from BL | -25 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | <30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | <0.5 | >1.23 |
| Phosphorus | mmol/L | | <0.8 | >1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | <18 | >32 |

# 11.7.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >160 |
| Diastolic Blood Pressure | mmHg | <45 | >100 |
| Heart Rate | bpm | <40 | >110 |

# 11.8. Appendix 8: Abbreviations & Trademarks

# 11.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ABC | Abacavir |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AGA | Appropriate for Gestational Age |
| A&R | Analysis and Reporting |
| APGAR | Appearance, Pulse rate, Grimace, Activity, Respiration |
| CDISC | Clinical Data Interchange Standards Consortium |
| CD4+ | Helper-inducer T-lymphocyte having surface antigen CD4 (cluster of differentiation 4) |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CSR | Clinical Study Report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| DAIDS | Division of AIDS |
| DBF | Database Freeze |
| DBR | Database Release |
| DTG | Dolutegravir |
| eCRF | Electronic Case Record Form |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FDC | Fixed Dose Combination |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library (GSK Standards Library) |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT(E) | Intent-To-Treat (Exposed) |
| IUGR | Intrauterine Growth Restriction |
| LGA | Large for Gestational Age |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| RAP | Reporting & Analysis Plan |
| RNA | Ribonucleic acid |
| SAC | Statistical Analysis Complete |
| SAS | Statistical Analysis Software |
| SDTM | Study Data Tabulation Model |
| SGA | Small for Gestational Age |

# 11.8.2. Trademarks

| Trademarks of the ViiV Healthcare | Trademarks not owned by the ViiV<br>Healthcare |
|---|---|
| Dolutegravir | SAS |
| Epzicom/Kivexa | WinNonlin |

### 11.9. Appendix 9: Final (End of Study) Analysis

This appendix provides the details of the planned analyses and data displays for the ING200336 final/End of Study (EoS) reporting. The primary analysis (i.e. interim analysis at 8-12 Weeks post-partum) was completed based on the original RAP. This appendix covers only analyses included in the final/EoS reporting and summarizes only the key endpoints of interest for the final analysis and summarizes any changes from the primary analysis. The details of the final/EoS reporting and analysis plan are described below:

- Analyses for which the data have not been changed since last interim analysis will
  not be reported to avoid redundancy. These reports include the analyses of
  demographic and baseline characteristics.
- 2. No subgroup analysis, hypotheses testing, or statistical analyses will be performed.
- 3. All required disclosure outputs following the FDAAA and EudraCT guidelines will be produced.
- 4. Pharmacokinetic, Virology and Maternal and Infant Outcome displays will not be produced in the EOS reporting effort.
- 5. Overview of the key endpoints for the study are below:
- Study Population:
  - Subject Disposition
  - Concomitant ART and non-ART Medications
  - Protocol Deviations
- Safety:
  - Extent of Exposure
  - Adverse Events
  - Maximum Post-Baseline Emergent Clinical Chemistry/ Haematology Toxicities/ Hepatobiliary Laboratory Abnormality Criteria
  - Positive Suicidal indication Alerts based on eC-SSRS
  - Summary of absolute values and change from baseline for Hematology and Chemistry parameters (as mentioned in Section 11.10.6)
- Efficacy:
  - Proportion of Subjects with Plasma HIV-1 RNA < 50 c/ mL observed data</li>
  - Change from Baseline in CD4+ cell count (cells/mm3) and Plasma HIV-1 RNA (log10 c/mL) by Visit
  - Absolute Values of Baseline and Post-baseline in CD4+ cell count (cells/mm3) by Visit
  - Incidence of disease progression and HIV- associated conditions

### 11.10. Appendix 10: List of Data Displays

All data displays will use the term "subject" rather than "participant" in accordance with CDSIC and GSK Statistical Display Standards.

### 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|--------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | NA |
| Efficacy | 2.1 to 2.n | NA |
| Safety | 3.1 to 3.n | NA |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Virology | 5.1 | NA |
| Maternal and Infant Assessment | 6.1 to 6.n | NA |
| Section | Listi | ngs |
| ICH Listings | 1 to | O X |
| Other Listings | y to | ) Z |

### 11.10.2. Mock Example Shell Referencing

Nonstandard specifications will be referenced as indicated and if required example mockup displays provided in Appendix 9: Example Mock Shells for Data Displays.

| Section | Table | Listing |
|-------------------|--------|---------|
| Pharmacokinetic | PK Tn | PK Ln |
| Maternal Outcomes | MAT Tn | MAT Ln |
| Infant Outcomes | INF Tn | INF Ln |
| Virology | VIR Tn | NA |

NOTES: For displays having Example shell as \*, refer to TANGO Study (Compound: GSK3515864, Study ID: 204862, Reporting Effort: primary 01)

### 11.10.3. Deliverables

| Delivery [Priority] | Description |
|---------------------|--------------------------------------------------|
| IA SAC | Interim Analysis Statistical Analysis Complete |
| EOS | Final End of Study Statistical Analysis Complete |

# 11.10.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | ITT-E | ES1 | Summary of Subject Disposition for the Subject Conclusion Record overall and by relationship to COVID-19 Pandemic | Table will be summarised overall and then by COVID-19 relationship | IA SAC, EOS |
| 1.2. | Enrolled | NS3 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | IA SAC |
| Demog | graphic and Bas | seline Characteris | tics | | |
| 1.3. | ITT-E | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | IA SAC |
| 1.4. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | IA SAC |
| 1.5. | ITT-E | DM6 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | IA SAC |

# 11.10.5. Efficacy Tables

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Plasma | HIV-1 RNA | | | | |
| 2.1 | ITT-E | * | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit | | IA SAC, EOS |
| 2.2 | ITT-E | * | Proportion of Subjects with Plasma HIV-1 RNA <400 c/mL by Visit | | IA SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3 | ITT-E | * | Summary of Change from Baseline in HIV-1 RNA (c/mL) by Visit | | IA SAC, EOS |
| CD4+ C | Cell Count | | | • | • |
| 2.4 | ITT-E | * | Summary of Change from Baseline in CD4+ Cell Count (cells/mm^3) by Visit | | IA SAC, EOS |
| 2.41 | ITT-E | * | Summary of Absolute Values of Baseline and Post-baseline in CD4+ Cell Count (cells/mm^3) by Visit | | IA SAC, EOS |
| Post- B | Post- Baseline Disease Progression | | | | |
| 2.5 | ITT-E | * | Summary of Post-Baseline HIV-1 Disease Progressions | | IA SAC, EOS |

# 11.10.6. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | e Events (AEs) | | | | |
| 3.1. | Safety | AE5B | Summary of All Adverse Events by System Organ Class,<br>Preferred term and Maximum Toxicity | Ct.gov | IA SAC, EOS |
| 3.2. | Safety | AE3 | Summary of Grade 2-4 Adverse Events by Overall Frequency | ICH E3 | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.3. | Safety | AE15 | Summary of Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT | IA SAC, EOS |
| 3.4. | Safety | AE3 | Summary of Non-Serious Drug-Related Adverse Events by Overall Frequency | Plain Language Summary requirements (PLS). | IA SAC, EOS |
| 3.5. | Safety | AE16 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Number of Subjects and<br>Occurrences) | FDAAA, EudraCT | IA SAC, EOS |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.6. | Safety | AE20 | Summary of Serious Fatal and Non-Fatal Drug-Related Adverse by Overall Frequency | Plain Language Summary requirements (PLS). | IA SAC, EOS |
| 3.7. | Safety | AE8 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | | IA SAC |
| 3.8. | Safety | * | Summary of Maximum Post-Baseline Emergent Chemistry Toxicities | The key parameters would include ALT, AST, Total bilirubin, serum creatinine and GFR | IA SAC, EOS |
| 3.9. | Safety | * | Summary of Maximum Post-Baseline Emergent<br>Hematology Toxicities | The parameters would include<br>Hemoglobin, platelets, WBC | IA SAC, EOS |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit | The key parameters would include ALT, AST, Total bilirubin, serum creatinine and GFR | IA SAC, EOS |
| 3.11. | Safety | LB1 | Summary of Hematology Changes from Baseline by Visit | The parameters would include Hemoglobin, platelets, WBC | IA SAC, EOS |
| 3.12. | Safety | LB1 | Summary of Urinalysis Changes from Baseline by Visit | Key parameters would be Urine protein/Creatinine ratio and Urine/Protein ratio | IA SAC |
| 3.13. | Safety | LB1 | Summary of Absolute Values of Chemistry for Baseline and Post-baseline by Visit | The key parameters would include ALT, AST, Total bilirubin, serum creatinine and GFR | IA SAC, EOS |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.14. | Safety | LB1 | Summary of Absolute Values of Hematology for Baseline and Post-baseline by Visit | The parameters would include Hemoglobin, platelets, WBC | IA SAC, EOS |

# 11.10.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| DTG P | DTG PK | | | | |
| 4.1. | PK | PK01 | Summary of Plasma DTG PK Concentration-Time Data by Visit and Nominal Time Relative to Dose | | IA SAC |
| 4.2. | PK | PK T1 | Summary of untransformed and loge-transformed Derived Plasma DTG PK Parameters | | IA SAC |

# 11.10.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| DTG P | ( | | | | |
| 4.1. | PK | PK24 | Individual Plasma DTG Concentration-Time Plots (linear and Semi-log) | | IA SAC |
| 4.2. | PK | PK17 | Mean Plasma DTG Concentration-Time plots (linear and semilog) | | IA SAC |
| 4.3. | PK | PK18 | Median Plasma DTG Concentration-Time plots (linear and semi-log) | | IA SAC |

# 11.10.9. Virology Tables

| Virology: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.1 | ITT-E | VIR T1 | Summary of Incidence of treatment-emergent genotypic and/or phenotypic resistance in subjects who meet confirmed virologic withdrawal criteria | | IA SAC |

### 11.10.10. Maternal and Infant Assessment Tables

| Maternal ar | Maternal and Infant Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Standard/<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.1 | Safety | MAT T1 | Summary of Maternal Outcomes | | IA SAC |
| 6.2 | Safety | INF T1 | Summary of Infant Outcomes at Birth | | IA SAC |

# 11.10.11. ICH Listings

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Standard /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | ITT-E | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | IA SAC, EOS |
| Protoc | ol Deviations | | | | |
| 2. | ITT-E | DV2 | Listing of Important Protocol Deviations | ICH E3 | IA SAC, EOS |
| 3. | ITT-E | DV2 | Listing of all non-Important COVID-19 related Protocol Deviations | | IA SAC, EOS |
| Demog | raphic and Base | line Characterist | ics | | • |
| 4. | ITT-E | DM2 | Listing of Demographic Characteristics | ICH E3 | IA SAC |
| 5. | ITT-E | DM9 | Listing of Race | ICH E3 | IA SAC |
| Exposi | Exposure and Treatment Compliance | | | | |
| 6. | ITT-E | EX3 | Listing of Investigational Product Exposure Data | ICH E3 | IA SAC, EOS |
| Advers | Adverse Events | | | | |
| 7. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | IA SAC, EOS |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Standard /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serious | s and Other Sign | ificant Adverse E | vents | | |
| 8. | Safety | AE8CPA | Listing of Non-Fatal Serious Adverse Events | ICH E3 | IA SAC |
| 9. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | IA SAC |
| 10. | Safety | AE8 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | ICH E3 | IA SAC, EOS |
| Labora | tory Assessment | ts | | | |
| 11. | Safety | LB5 | Listing of Clinical Chemistry Laboratory Data | ICH E3 | IA SAC, EOS |
| 12. | Safety | LB5 | Listing of Haematology Laboratory Data | ICH E3 | IA SAC, EOS |
| 13. | Safety | UR2 | Listing of Urinalysis Data | ICH E3 | IA SAC, EOS |

# 11.10.12. Non-ICH Listings

| Non-ICH: Listings | | | | |
|---|---|---|---|---|
| No. | No. Population Example Shell Title Programming Notes Deliverable [Priority] | | | |
| Prior and Concomitant Medications | | | | |
| 14. | ITT-E | CM3 | Listing of Concomitant Non-ART Medications | IA SAC, EOS |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 15. | ITT-E | CM3 | Listing of Concomitant ART Medications | | IA SAC, EOS |
| 16. | ITT-E | * | Listing of Relationship Between ATC Level 1, Ingredient and Verbatim Text | | IA SAC, EOS |
| 17. | ITT-E | * | Listing of Relationship Between ATC Level 4, Ingredient and Verbatim Text | | IA SAC, EOS |
| Adverse E | Events | | | | |
| 18. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | IA SAC |
| Pandemic | | | | | |
| 19. | Safety | PAN12 | Listing of COVID-19 Assessments and Symptom assessments | | IA SAC, EOS |

| Non-ICH: | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Non-Lab | Non-Laboratory values | | | | |
| 20. | Safety | ECSSRS4 | Listing of C-SSRS Suicidal Ideation and Behaviour Data | | IA SAC, EOS |
| Subject D | Disposition | | | | • |
| 21. | ITT-E | * | Listing of Investigational Product Accountability | | IA SAC, EOS |
| 22. | ITT-E | TA1 | Listing of Planned and Actual Treatments | | |
| 23. | All Subjects<br>Screened | * | Listing of Study Populations | | IA SAC |
| 24. | Enrolled | * | Listing of Subject Recruitment by Country and Site Number | Add a column "ARIA-ING117172<br>Unique Subject ID" | IA SAC |
| 25. | ITT-E | * | Listing of Visit Dates | | IA SAC, EOS |
| 26. | ITT-E | CDC3 | Listing of CDC Classification of HIV Infection at Baseline | | IA SAC |
| 27. | ITT-E | RF2 | Listing of HIV Risk Factors | | IA SAC |
| Medical C | Conditions | | | | |
| 28. | ITT-E | MH2 | Listing of Current and Past Medical Conditions at Baseline | | IA SAC |
| Baseline | Characteristic | s | - | | |
| 29. | ITT-E | * | Listing of Baseline Cardiovascular Risk Assessment Data | | IA SAC |
| 30. | ITT-E | * | Listing of History of Cardiac Therapeutic Procedures | | IA SAC |
| 31. | ITT-E | * | Listing of Cardiovascular Events at Baseline | | IA SAC |
| 32. | ITT-E | MAT L2 | Listing of Maternal History | | IA SAC |
| Efficacy | | | | | |
| 33. | ITT-E | * | Listing of Quantitative Plasma HIV-1 RNA | | IA SAC, EOS |

| Non-ICH: | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 34. | ITT-E | * | Listing of CD4+ Cell Count Data | | IA SAC, EOS |
| Vital Sign | s | | | | |
| 35. | Safety | VS4 | Listing of All Vital Signs Data | | IA SAC, EOS |
| PK Endpo | ints | | | | |
| 36. | PK | PK L1 | Listing of Plasma DTG PK Concentration-Time Data | | IA SAC |
| 37. | PK | PK L2 | Listing of Plasma DTG PK Parameters | | IA SAC |
| Maternal a | Maternal and Infant Endpoints | | | | |
| 38. | Safety | MAT L1 | Listing of Maternal Outcomes | | IA SAC |
| 39. | Safety | MAT L3 | Listing of Pregnancy Risk Assessment | | IA SAC |
| 40. | Safety | INF L1 | Listing of Infant Outcomes | | IA SAC |

# 11.11. Appendix 11: Example Mock Shells for Data Displays

Example mock shells for Data Displays will be provided in a separate document.

#### ViiV Healthcare group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for ING200336: A Prospective, Interventional Pharmacokinetic and Safety Study of DTG/ABC/3TC in Pregnant Women |
|---|---|---|
| <b>Compound Number</b> | : | GSK1349572+GR109714+GI265235 (GSK2619619) |
| Clinical Study<br>Identifier | : | ING200336 |
| Effective Date | : | 03-MAR-2021 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 200336.
- This RAP is intended to describe all the planned analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverables.

### RAP Author(s):

| Author | Date |
|------------------------------------|-------------|
| Lead | |
| PPD | 17 FED 2021 |
| Junior Statistician, Biostatistics | 17-FEB-2021 |

Copyright 2021 ViiV Healthcare group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

### **RAP Team Reviews:**

### **RAP Team Review Confirmations**

(Method: E-mail)

| Reviewer | Date |
|---------------------------------------------------|--------------|
| PPD | 25 EED 2021 |
| Principal Statistician, Biostatistics, GSK | 25-FEB-2021 |
| PPD | 25 FED 2021 |
| Principal Programmer/ Analyst, Biostatistics, GSK | 25-FEB-2021 |
| PPD | 01.14.0.2021 |
| PPD , ViiV | 01-MAR-2021 |
| PPD | |
| Manager, Clinical Pharmacology | 01-MAR-2021 |
| CPMS, GSK | |
| PPD | |
| , Global Clinical Safety and | 25-FEB-2021 |
| Pharmacovigilance, GSK | |
| PPD | 25-FEB-2021 |
| Clinical Development Leader, ViiV | 23-FED-2021 |
| PPD | |
| Discovery Medicine Lead, N6LS | 25-FEB-2021 |
| ViiV | |
| PPD | 25-FEB-2021 |
| Clinical Data Analyst, GSK | 23-FED-2021 |

# **Clinical Statistics and Clinical Programming Line Approvals:**

# Approved through email by:

| Approv | er | Date | |
|-------------|---------------|------|-------------|
| PPD Manager | r, Statistics | | 03-MAR-2021 |
| PPD | | | 02-MAR-2021 |
| PPD | Programming | | 02-MAK-2021 |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRODUCT | TON | 6 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | | |
| ۷. | | ges to the Protocol Defined Statistical Analysis Plan | |
| | | Objectives and Endpoints | |
| | | tical Hypotheses / Statistical Analyses | |
| | | · | |
| | | n AnalysesAnalyses | |
| | 2.0. Fillal I | Analyses | 9 |
| 3. | ANALYSIS P | OPULATIONS | 11 |
| ٠. | | col Deviations | |
| 4. | | ATIONS FOR DATA ANALYSES AND DATA HANDLING | 40 |
| | | NS | |
| | 4.1. Study | Treatment & Sub-group Display Descriptors | 12 |
| | | ine Definitions | |
| | | centre Studies | |
| | | ination of Covariates, Other Strata and Subgroups Considerations for Data Analyses and Data Handling | 12 |
| | | entionsentions for Data Arialyses and Data Handling | 12 |
| 5. | STUDY POP | ULATION ANALYSES | 14 |
| | 5.1. Overv | view of Planned Study Population Analyses | 14 |
| 6. | EFFICACY A | NALYSES | 16 |
| 0. | | oint / Variables | |
| | | nary Measure | |
| | | ation of Interest | |
| | | egy for Intercurrent (Post-Randomization) Events | |
| | | cy Analyses / Methods | |
| | | -,, | |
| 7. | | ALYSES | |
| | | se Events Analyses | |
| | 7.2. Clinica | al Laboratory and Other Safety Analyses | 19 |
| 8. | PHARMACO | KINETIC ANALYSES | 20 |
| ٥. | | ary and Secondary Pharmacokinetic Analyses | |
| | 8.1.1. | · | |
| | 0 | 8.1.1.1. Drug Concentration Measures | |
| | | 8.1.1.2. Derived Pharmacokinetic Parameters | |
| | 8.1.2. | | |
| | 8.1.3. | • | |
| | 8.1.4. | • | |
| | 8.1.5. | | |
| | | • | |
| 9 | MATERNAL | AND INFANT ANALYSES | 22 |

| | 9.1. | Maternal | l Outcomes | <mark>22</mark> |
|---|---|---|---|---|
| | | 9.1.1. | Endpoints/Variables | <mark>22</mark> |
| | | 9.1.2. | Summary Measure | <mark>22</mark> |
| | | 9.1.3. | Population of Interest | |
| | | 9.1.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 9.1.5. | Statistical Analyses/ Methods | |
| | 9.2. | | utcomes | |
| | | 9.2.1. | Endpoints/Variables | |
| | | 9.2.2. | Summary Measure | |
| | | 9.2.3. | Population of Interest | |
| | | 9.2.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 9.2.5. | Statistical Analyses/ Methods | 24 |
| 10. | VIROL | OGY ANA | ALYSIS | 25 |
| | | 10.1.1. | | |
| | | 10.1.2. | | |
| | | 10.1.3. | | |
| 11. | | | x 1: Schedule of Activities | |
| | 11.1. | | Protocol Defined Schedule of Events | |
| | 11.2. | | x 2: Assessment Windows | |
| | 11.2. | 11.2.1. | Definitions of Assessment Windows for Analyses | |
| | | 11.2.1. | Definitions of Assessment Windows for Inclusion in the PK | 23 |
| | | 11.2.2. | Analysis | 30 |
| | | 11.2.3. | Stages of Pregnancy used for Pharmacokinetics | |
| | | 11.2.4. | | |
| | 11.3. | | x 3: Study Phases and Treatment Emergent Adverse | |
| | | | | 31 |
| | | 11.3.1. | Study Phases | |
| | | | 11.3.1.1. Treatment States for Laboratory, HIV | |
| | | | Associated Conditions, Vital Signs, and | |
| | | | Genotypic and Phenotypic Data | 31 |
| | | | 11.3.1.2. Treatment States for Prior/Concomitant/Post- | |
| | | | Therapy Medications Data | 31 |
| | | | 11.3.1.3. Treatment States for AE Data | |
| | | 11.3.2. | Treatment Emergent Flag for Adverse Events | |
| | 11.4. | | x 4: Data Display Standards & Handling Conventions | |
| | | 11.4.1. | Reporting Process | |
| | | 11.4.2. | Reporting Standards | |
| | | 11.4.3. | Reporting Standards for Pharmacokinetic | |
| | 11.5. | | x 5: Derived and Transformed Data | |
| | | 11.5.1. | General | |
| | | 11.5.2. | Study Population | |
| | | 11.5.3. | Efficacy | |
| | | 11.5.4. | Safety | |
| | 44.0 | 11.5.5. | Pharmacokinetic | |
| | 11.6. | | x 6: Reporting Standards for Missing Data | |
| | | 11.6.1. | Premature Withdrawals | |
| | | 11.6.2. | Handling of Missing Data | |
| | 117 | Annord: | 11.6.2.1. Handling of Missing and Partial Datesx 7: Values of Potential Clinical Importance | |
| | 11./. | ADDELIGI | x /. values ui fuleiiliai Ciiilicai IIIIDUI laiice | |

# 2021N493381\_00 ING200336

| | 11.7.1. | Laboratory Values | 41 |
|--------|----------|-------------------------------------------|-----------|
| | 11.7.2. | Vital Signs | 41 |
| 11.8. | | c 8: Abbreviations & Trademarks | |
| | 11.8.1. | Abbreviations | 42 |
| | 11.8.2. | Trademarks | 43 |
| 11.9. | Appendix | c 9: List of Data Displays | 44 |
| | 11.9.1. | Data Display Numbering | 44 |
| | 11.9.2. | Mock Example Shell Referencing | 44 |
| | 11.9.3. | Deliverables | 44 |
| | 11.9.4. | Study Population Tables | 45 |
| | 11.9.5. | Efficacy Tables | 45 |
| | 11.9.6. | Safety Tables | 46 |
| | 11.9.7. | Pharmacokinetic Tables | <b>50</b> |
| | 11.9.8. | Pharmacokinetic Figures | 51 |
| | | Virology Tables | |
| | 11.9.10. | Maternal and Infant Assessment Tables | 52 |
| | 11.9.11. | ICH Listings | 53 |
| | | Non-ICH Listings | |
| 11.10. | | 10: Example Mock Shells for Data Displays | |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol: 200336

| Revision Chronology: | | |
|------------------------|-------------|-------------------|
| GlaxoSmithKline Date | | Version |
| <b>Document Number</b> | | |
| 2013N166290 00 | 18-DEC-2013 | Original |
| 2013N166290 01 | 15-APR-2014 | Amendment No.: 01 |
| 2013N166290 02 | 23-APR-2014 | Amendment No.: 02 |
| 2013N166290 03 | 19-JUN-2018 | Amendment No.: 03 |

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

### 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Pharmacokinetic Analysis: Log-transformed PK parameters except tmax will be analysed by analysis of variance | No ANOVA will be done. | Very few subjects<br>will be recruited |
| <ul> <li>Efficacy Endpoints for Infants:</li> <li>Proportion of subjects with plasma HIV-1 RNA &lt; 50 c/mL and &lt;400 c/mL over time.</li> <li>Absolute values and changes from Baseline in CD4+ T cell counts over time.</li> <li>Incidence of disease progression (HIV-associated conditions, acquired immunodeficiency syndrome [AIDS] and death).</li> </ul> | These data were not collected for Infants. | Inconsistencies within the protocol. The data for these endpoints were not collected in infants. |

# 2.2. Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Mother | |
| To describe the total plasma DTG PK parameters with the DTG/ABC/3TC FDC during Weeks 18-26, Weeks 30 – 36 of the third trimester of the pregnancy and 8-12 weeks postpartum | <ul> <li>Area under the concentration-time curve<br/>during a 24-hour interval at steady state<br/>[AUC24], maximal drug concentration<br/>[Cmax], drug concentration at the end of<br/>dosing interval [Cτ], Tmax, C0,<br/>apparent clearance [CL/F[, steady state<br/>volume of distribution [Vss/F] and the<br/>half-life [t½]) of DTG</li> </ul> |
| To further characterize the safety and tolerability of DTG/ABC/3TC FDC when used during pregnancy | <ul> <li>Incidence and severity of AEs and laboratory abnormalities.</li> <li>Absolute values and changes over time in laboratory parameters;</li> <li>Proportion of subjects who discontinue treatment due to AEs;</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| M | other |
| To assess the antiviral activity of the DTG/ABC/3TC FDC when administered during pregnancy To assess the immunologic activity of | <ul> <li>Absolute values and change from<br/>Baseline HIV1 RNA over time.</li> <li>Proportion of subjects with plasma HIV-<br/>1 RNA &lt;50 and &lt;400 c/mL over time</li> <li>Absolute values and change from</li> </ul> |
| DTG/ABC/3TC FDC • Incidence of disease progression | Baseline in CD4+ cell count over time. HIV-associated conditions, acquired immunodeficiency syndrome [AIDS] and death |
| To assess the incidence of treatment – emergent genotypic and phenotypic resistance in subjects who meet virologic withdrawal criteria | Treatment-emergent genotypic and<br>phenotypic resistance in subjects who<br>meet confirmed virologic withdrawal<br>criteria |
| To evaluate the unbound DTG concentrations in plasma during Weeks 18-26 and Weeks 30-36 of the pregnancy and 8-12 weeks postpartum | Unbound concentrations and Unbound<br>fraction at 3 and 24 hours post dose in<br>the third trimester and postpartum. |
| To compare the DTG concentrations<br>in plasma from cord blood with those<br>in maternal plasma at the time of<br>delivery | Total DTG concentrations in plasma<br>from cord blood and those in maternal<br>plasma at the time of delivery. |
| To characterize pregnancy (maternal) outcomes | Pregnancy outcomes; Pregnancy risks |

| Objectives | Endpoints |
|---|---|
| To characterize birth outcomes | <ul> <li>Birth outcomes (per pregnancy outcomes endpoint above)</li> </ul> |
| Infa | ant |
| To characterize infant outcomes at birth | Infant outcomes at birth |
| To characterize the safety of<br>DTG/ABC/3TC FDC to the<br>developing fetus | <ul> <li>Proportion of pregnancies with and<br/>without demonstrated congenital<br/>malformations</li> </ul> |

### 2.3. Study Design

| Overview of St | Overview of Study Design and Key Features |
|---|---|
| Design<br>Features | <ul> <li>This is a single arm open-label interventional study for women who<br/>become pregnant while participating in ING117172 on the<br/>DTG/ABC/3TC FDC treatment arm.</li> </ul> |
| Dosing | <ul> <li>All subjects will be administered DTG 50 mg/ABC 600 mg/3TC 300<br/>mg FDC tablet administered once daily.</li> </ul> |
| Time & Events | • [Refer to Appendix 1: Schedule of Activities] |
| Treatment<br>Assignment | <ul> <li>Subjects will initiate therapy with DTG/ABC/3TC FDC following<br/>confirmation of fulfilment of study entry criteria. A unique treatment<br/>number will be assigned for each subject participating in the study.<br/>Subjects who are enrolled into the trial and subsequently withdrawn<br/>may not be re-screened.</li> </ul> |
| Interim<br>Analysis | <ul> <li>No interim analysis was planned, however protocol allowed further<br/>data cuts and analyses to be conducted as necessary to support<br/>regulatory requests, submissions and/or publications. The study<br/>recruitment was terminated early which triggered reporting of the<br/>primary endpoint.</li> </ul> |

### 2.4. Statistical Hypotheses / Statistical Analyses

This is a single arm open-label interventional study for women who become pregnant while participating in ING117172. No formal hypotheses testing will be performed.

### 2.5. Interim Analyses

No interim analyses were formally planned, however the protocol allows further data cuts and analyses are conducted as necessary to support regulatory requests, submissions and/or publications. The planned analyses will be performed after the completion of the following sequential steps:

- 1. Subjects are considered to have completed the study after completing the postpartum evaluation approximately 8-12 weeks post-delivery. The primary outcome analyses will take place after the last subject enrolled gives birth and completes their last visit.
- 2. All required database cleaning activities have been completed.

### 2.6. Final Analyses

Subjects may continue to receive DTG/ABC/3TC FDC after completion of the primary endpoint assessments, until study medications are locally approved and commercially available (or they meet a criteria for withdrawal). During this time, subjects will be monitored every 12 weeks to ensure they continue to derive clinical benefit from DTG/ABC/3TC FDC.

A final End-of-Study analysis will be conducted when all subjects have completed the study and final database release (DBR), source data lock (SDL) and database freeze (DBF) have been declared by Data Management.

# 3. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All subjects<br>Screened | All participants who were screened for eligibility | Study Population |
| Enrolled | All participants who passed screening and entered the study | Study Population |
| Safety/ITT-E | All participants who received at least one dose of study treatment. | <ul><li>Study Population</li><li>Safety</li><li>Efficacy</li></ul> |
| Pharmacokinetic<br>(PK) | All participants in the Safety population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as missing values) | • PK |
| | Note: PK samples that may be affected by protocol<br>deviations will be reviewed by the study team to<br>determine whether or not the sample will be excluded. | |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

### 3.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) and non-important COVID-19 related protocol deviations will be listed.

# 4. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

### 4.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | Data Displays for Reporting | | |
| Code Description Description Orde | | Order | |
| Α | DTG/ABC/3TC FDC once daily | DTG/ABC/3TC | 1 |

No subgroup analysis will be done.

#### 4.2. Baseline Definitions

For all endpoints (unless otherwise stated) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data are missing no derivation will be performed and baseline will be set to missing.

Unless otherwise specified, the baseline definitions specified in the table below will be used for derivations for endpoints/parameters and indicated on listings.

| Definition | Reporting Details |
|------------------------|-----------------------------------------------------|
| Change from Baseline | Post-Dose Visit Value Baseline |
| % Change from Baseline | 100 x [(Post-Dose Visit Value Baseline) / Baseline] |

#### 4.3. Multicentre Studies

There are no planned adjustments made for multiple centres in this study.

# 4.4. Examination of Covariates, Other Strata and Subgroups

No covariates, Strata or Subgroups will be considered for descriptive summaries or Statistical analysis.

# 4.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:
| Section | Component |
|---------|----------------------------------------------------------------|
| 11.2 | Appendix 2 : Assessment Windows |
| 11.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Reporting Standards for Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |

### 5. STUDY POPULATION ANALYSES

### 5.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Enrolled and ITT-E population.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 9: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data Display | y's Generated |
|---|---|---|
| | Table | Listing |
| Randomisation | | • |
| Randomisation | | Y |
| Subject Disposition | | |
| Study Populations | | Υ |
| Subject Recruitment by country and site ID | Y | Y |
| Disposition (overall and by relationship to COVID-19 Pandemic) | Υ | |
| Reasons for Withdrawal | | Y |
| Study Visit Dates | | Υ |
| Protocol Deviations | | |
| Important Protocol Deviations | | Υ |
| Non-Important COVID-19 related Protocol Deviations | | Υ |
| <b>Demography and Baseline Characteristics</b> | | |
| Demographic Characteristics | Y | Υ |
| Age Ranges | Y | |
| Race | Y | Υ |
| CDC Classification of HIV infection at Baseline | | Υ |
| Cardiovascular Risk Assessments at Baseline | | Υ |
| History of Cardiac Therapeutic Procedures | | Υ |
| Cardiovascular Events at Baseline | | Υ |
| Maternal History (Pregnancy History) | | Y |
| Medical Conditions, Concomitant Medications & Ant | iretroviral Therapy | |
| Medical Conditions (Current and Past) | | Y |
| Concomitant Medications (non-ART) | | <b>Y</b> [1] |
| Prior and Concomitant ART Medications | | <b>Y</b> [2] |

| Display Type | Data Display's Generated | |
|-------------------------|--------------------------|---|
| | Table Listing | |
| Other | | |
| Investigational Product | | Y |

#### **Notes:**

- Y = Display Generated
- 1. One listing for concomitant non-ART medications and one listing showing the relationship between verbatim text, ingredient and ATC Level 1.
- 2. One listing for Prior ART, one listing for concomitant ART and one listing showing the relationship between verbatim text, ingredient, combination and ATC Level 4.

#### 6. EFFICACY ANALYSES

#### 6.1. Endpoint / Variables

#### Mother

- Absolute value and change from baseline in HIV-1 RNA over time
- Proportion of subjects with plasma HIV-1 RNA <50 and <400 c/mL over time</li>
- Absolute value and change from baseline in CD4+ Cell count over time
- Disease progression and HIV associated conditions

#### 6.2. Summary Measure

Efficacy data will be presented in tabular form and will be summarized descriptively by visit.

#### 6.3. Population of Interest

The efficacy analyses will be based on the Intent-To-Treat- Exposed population, unless otherwise specified.

#### 6.4. Strategy for Intercurrent (Post-Randomization) Events

Not applicable.

### 6.5. Efficacy Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 6.1 will be listed and summarised.

Table 3 Overview of Planned Efficacy Analyses

| Endpoints | Absolute | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sumr | mary | Indiv | idual | Sumr | Summary | | ividual |
| | T | F | F | L | Т | F | F | L |
| Quantitative Plasma H | IIV-1 RNA | | | | | | | |
| Observed over time | | | | Υ | Y | | | |
| Proportion of<br>Subjects with Plasma<br>HIV-1 RNA <400<br>copies/mL | Y | | | | | | | |
| Proportion of<br>Subjects with Plasma | Y | | | | | | | |

| Endpoints | Absolute | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sumr | mary | Indiv | idual | Sumr | mary | Individual | |
| | Т | F | F | L | Т | F | F | L |
| HIV-1 RNA <50<br>copies/mL | | | | | | | | |
| CD4+ Cell Count | | | | | | | | |
| Observed over time | | | | Υ | Y | | | |
| Post-baseline HIV-1 Disc | ease Progr | ession | | | | | | |
| Incidence of<br>disease<br>progression <sup>[1]</sup> | Y | | | | | | | |

**NOTES:** L = Listing, Y = Yes display generated.

<sup>1.</sup> HIV-associated conditions, acquired immunodeficiency syndrome [AIDS] and death

### 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

### 7.1. Adverse Events Analyses

The details of the planned displays are provided in Appendix 9: List of Data Displays.

Table 4 Overview of Planned Safety Analyses

| | A | bsolute |
|---|---|---|
| Display Type | Summary | Individual |
| | T | L |
| Exposure Data | | Y |
| All Adverse Events | | Y |
| Non-Fatal serious Adverse<br>Events | | Y |
| Non-Serious Drug-Related<br>Adverse Events by Overall<br>Frequency | Y | |
| All Adverse Events by System<br>Organ Class, Preferred Term and<br>Maximum Toxicity | Y | |
| Non-serious Adverse Events by<br>System Organ Class and<br>Preferred Term (Number of<br>Subjects and Occurrences) | Y | |
| Grade 2-4 Adverse Events by<br>Overall Frequency | Y | |
| Serious Adverse Events by<br>System Organ Class and<br>Preferred Term (Number of<br>Subjects and Occurrences) | Y | |
| Serious Fatal and Non-Fatal<br>Drug-Related Adverse Events by<br>Overall Frequency | Y | |

| | A | bsolute |
|---|---|---|
| Display Type | Summary | Individual |
| | Т | L |
| Reasons for Considering as a<br>Serious Adverse Event | | Y |
| Adverse Events Leading to<br>Permanent Discontinuation of<br>Study Treatment or Withdrawal<br>from Study | Y | Y |
| Relationship of Adverse Event<br>System Organ Classes, Preferred<br>Terms, and Verbatim Text | | Y |
| COVID-19 Assessments and Symptom assessments | | Y |

**NOTES:** • T = Table, L = Listing, Y = Yes display generated.

### 7.2. Clinical Laboratory and Other Safety Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests and Urinalysis, and non-laboratory safety test results including vital signs, cardiovascular events and suicidality monitoring tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 9: List of Data Displays.

| Endpoint | | Abs | solute | | С | Change from Baseline | | | | Max Post BL | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indi | vidual | Stats | Analys | nalysis Summary | | nary | Summary | | y |
| | T | F | F | L | T | F | L | T | F | Т | F | L |
| Laboratory values | | | | | | | | | | | | |
| Clinical Chemistry | | | | Y | | | | Υ | | Υ | | |
| Haematology | | | | Y | | | | Y | | Υ | | |
| Urinalysis | | | | Υ | | | | Υ | | | | |
| Non-Laboratory va | lues | | | | | | | | | | | |
| Vital Signs | | | | Υ | | | | | | | | |
| Suicidal Ideation | | | | Υ | | | | | | | | |
| and Behaviour | | | | | | | | | | | | |
| Data | | | | | | | | | | | | |
| Others | | | | | | | | | | | | |
| COVID-19 | | | | Υ | | | | | | | | |
| Symptom and | | | | | | | | | | | | |
| assessments | | | | | | | | | | | | |

**NOTES**: T=Table, F=Figure, L = Listing, Y = Yes display generated

#### 8. PHARMACOKINETIC ANALYSES

#### 8.1. Primary and Secondary Pharmacokinetic Analyses

#### 8.1.1. Endpoint / Variables

Pharmacokinetic parameters will be determined from the plasma concentration-time data, as data permits.

#### **Primary PK Analysis Endpoints:**

DTG AUC(0- $\tau$ ), Cmax, C $\tau$ , CL/F, Vss/F, and  $t_2$  based on intensive PK sampling during the second and third trimesters of pregnancy (Weeks 18-26 and 30-36) and at 8-12 weeks postpartum will be determined, as data permits.

#### **Secondary PK Analysis Endpoints**

- C0 and Tmax based on intensive PK sampling during the second and third trimesters of pregnancy (Weeks 18-26 and 30-36) and at 8-12 weeks postpartum
- C3h,u and C24h,u and fu at the PK visits during the second and third trimesters and at 8-12 weeks postpartum
- Total DTG concentrations in plasma from cord blood compared to those in maternal plasma at the time of delivery.

#### 8.1.1.1. Drug Concentration Measures

All PK concentration summary and listing displays will be based on Pharmacokinetic population. Concentrations of DTG in plasma will be listed and summarized according to GSK standards, where applicable (Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Standards for Pharmacokinetic).

DTG concentration listings for the PK population will be sorted by subject and time relative to dose, noting the study visit; summaries will be presented by time relative to dose at each PK visit -Weeks 18-26 and Weeks 30-36 of pregnancy, and at 8-12 weeks post-partum (See Appendix 2: Section 11.2.3 for details). At each PK visit, samples will be collected prior to dosing and at 1,2, 3, 4, 6, 8, 12 and 24 hours post dosing. The predose sample should be collected within 15 minutes prior to the dose on the day of PK visit. DTG concentrations in plasma from cord blood will also be collected at the time of delivery will be compared with those in maternal plasma at the time of delivery.

#### 8.1.1.2. Derived Pharmacokinetic Parameters

PK analysis will be the responsibility of the Clinical PK Modeling & Simulation department within GlaxoSmithKline. Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 5.2 or higher. All calculations of non-

compartmental parameters will be based on actual sampling times recorded during the study. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

Table 5 Table of Derived PK Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | DTG Area under the plasma concentration time curve at steady state during a dosing interval |
| C0 | DTG Pre-dose plasma concentration |
| Cmax | DTG maximum observed plasma concentration determined directly from the concentration-time data. |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Сτ | Drug concentration at the end of dosing interval. |
| CL/F | Apparent oral clearance. |
| Vss/F | Apparent volume of distribution after extravascular (e.g., oral) administration. |
| t½ | DTG half-life. |
| C3h,u | Unbound DTG concentration in plasma at 3 hours post dose |
| C24h, u | Unbound DTG concentration in plasma 24 hours post dose |
| Weight Normalised CL/F | Apparent oral clearance |
| Weight Normalised<br>Vss/F | Apparent volume of distribution after extravascular (e.g., oral) administration |
| fu3h and fu24h | Unbound fraction at 3 hours and 24 hours post dose, calculated as: |
| | fu Cunbound/Ctotal |
| | where Cunbound and Ctotal are the unbound and total concentration of DTG in plasma, respectively. |

#### 8.1.2. Summary Measure

Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively by time relative to dose at each PK visit -Weeks 18-26 and Weeks 30-36 of pregnancy, and at 8-12 weeks post-partum (See Appendix 2: Section 11.2.3 for details).

#### 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

#### 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

Not Applicable.

#### 8.1.5. Statistical Analyses / Methods

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

Table 6 provides an overview of the planned analyses, with full details being presented in Appendix 9: List of Data Displays.

Table 6 Overview of Planned Pharmacokinetic Analyses

| | | Untrar | sforme | i | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| <b>End Point</b> | Summary | | Individual | | Summary | | Individual | |
| | T | F | F | L | T | F | F | L |
| PK Concentrati | PK Concentrations | | | | | | | |
| Plasma DTG<br>Concentrations | Y | Y | Y | Y | Y | Y | Y | |
| PK Parameters | | | | | | | | |
| Plasma DTG<br>Parameters | Y | | | Y | Y | | | |

Note: T Table, F Figure, L Listing, Y = Yes display generated

#### 9. MATERNAL AND INFANT ANALYSES

#### 9.1. Maternal Outcomes

#### 9.1.1. Endpoints/Variables

- Pregnancy outcomes variables: Spontaneous loss/miscarriage, Elective termination, Still birth, Live birth. In case of Live birth applicable Birth outcome categories will be listed.
- Maternal History
- Previous and Current Pregnancy risk assessment

#### 9.1.2. Summary Measure

Current Maternal data will be summarised over each maternal outcome.

#### 9.1.3. Population of Interest

The Maternal Outcome analysis will be based on the Safety population, unless otherwise specified.

#### 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

Not applicable.

#### 9.1.5. Statistical Analyses/ Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, all endpoints / variables defined in Section 9.1.1 will be listed. The pregnancy outcomes will be summarised.

#### 9.2. Infant Outcomes

#### 9.2.1. Endpoints/Variables

Infant outcome variables:

- Infant gestational age,
- Gestational length,
- Gestational weight (including percentiles, SGA, AGA, LGA, IUGR [IUGR in case of SGA only])
- Head circumference
- APGAR (Appearance, Pulse Rate, Grimace Reflex, Activity, Respiration) one and five minute scores
- Presence or absence of major congenital abnormalities at birth.
- HIV Status of Infant at 8-12 week postpartum visit

#### 9.2.2. Summary Measure

The Infant data will be summarised over each outcome.

#### 9.2.3. Population of Interest

The Infant Outcome analysis will be based on the Safety Population, unless otherwise specified.

#### 9.2.4. Strategy for Intercurrent (Post-Randomization) Events

Not applicable.

### 9.2.5. Statistical Analyses/ Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.2.1 will be listed and summarised.

### 10. VIROLOGY ANALYSIS

#### 10.1.1. Endpoints/Variables

Treatment-emergent genotypic and phenotypic resistance in subjects who meet confirmed virologic withdrawal criteria

#### 10.1.2. Population of Interest

The virology analyses will be based on the ITT-E population, unless otherwise specified.

### 10.1.3. Statistical Analyses/Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoint defined in Section 10.1.1 will be summarised.

### 11. APPENDICES

### 11.1. Appendix 1: Schedule of Activities

### 11.1.1. Protocol Defined Schedule of Events

| Procedures | Screen'." | Day 1 | Ante partum | Delivery | Post-Partum | Continuation<br>Phase | Withdrawal | Follow-up <sup>12</sup> |
|---|---|---|---|---|---|---|---|---|
| | | | Monthly – every 4<br>weeks | | 8-12 weeks<br>post delivery | Every 12 weeks<br>after Post<br>Partum Visit | | |
| Written Informed Consent | X | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | X | | | | | | |
| Subject Demography | X | | | | | | | |
| Medical History <sup>1</sup> | | X | | | X | X | | |
| Concurrent medical conditions | | X | | | | | | |
| CDC HIV-1 classification | | X | | | | | | |
| HIV-associated conditions | | | X | X | X | X | X | X |
| Cardiovascular risk<br>assessment <sup>2</sup> | * | | | | | | | |
| Prior Art history | ± | | | | | | | |
| Gravidity Maternal history | | X | | | | | | |
| Pregnancy risk assessment | X | X | X | | | | | |
| Uteroplacental Outcomes<br>at Delivery <sup>a</sup> | | | | X | | | | |
| Infant Outcomes4 | | | | X | X | X | | X |
| Concomitant Medication | Х | Х | X | X | X | Х | Х | X |
| Limited Physical<br>Examination <sup>6</sup> | | X | X | | X | X | Х | X |
| Adverse Events | X | X | X | X | X | X | X | X |

| Procedures | Screen'." | Day 1 | Ante partum | Delivery | Post-Partum | Continuation<br>Phase | Withdrawal | Follow-up <sup>12</sup> |
|---|---|---|---|---|---|---|---|---|
| | | | Monthly – every 4<br>weeks | | 8-12 weeks<br>post delivery | Every 12 weeks<br>after Post<br>Partum Visit | | |
| Serious Adverse Events® | X | X | X | <b>X</b> 6 | Х | X | X | X |
| Pharmacokinetic<br>Sampling <sup>7</sup> | | | Χε | X | X | | | |
| Cord & maternal blood<br>sample <sup>8</sup> | | | | X | | | | |
| Columbia Suicidality<br>Severity Rating Scale | | X | X | | X | X | X | |
| Laboratory Assessments | | | | | | | | |
| Pregnancy Assessment | | X | | | Х | X | | |
| Hematology | ** | ** | X | | Х | Х | X | X |
| Clinical Chemistry | ** | ** | X | | X | X | X | X |
| Urinalysis. Including | ** | | X | | X | X | | X |
| dipstick for protein<br>analysis | | | | | | | | |
| Quantitative plasma HIV-1<br>RNA <sup>10</sup> | ** | ** | X | X | X | X | X | |
| Lymphocyte subsets | ** | ** | X | <b>X</b> 6 | X | X | | X |
| PGx Sampling <sup>11</sup> | | X | | | | | | |
| Plasma for storage12 | X | X | X | X | X | X | X | X |
| Dispense IP | | X | X | X | X | Х11 | | |

<sup>\*</sup>Baseline information, including cardiovascular risk and prior ART therapy will be transferred from ING117172 to serve as baseline/screening data in this study.

- 1. Medical History includes any changes in smoking status
- 2. Assessment for cardiovascular risk will include height, weight, blood pressure, smoking history, medical conditions and will have previously been collected in ING117172
- 3. Assessment of pregnancy outcomes (e.g., spontaneous losses, induced abortions, still births, pre-term births, preeclampsia)
- 4. Assessment of maternal and infant outcomes, including live births, gestational age, presence or absence of major congenital abnormalities, and infant height, weight, [including percentiles, SGA, AGA, LGA, IUGR], head circumference, and presence or absence of major congenital abnormalities at birth. If known, HIV status of the infant will be collected at the 8-12 week post-partum visit.
- 5. Limited physical examination to include blood pressure at Baseline (recorded in eCRF), heart rate and weight at each visit (recorded in eCRF at Baseline and on lab requisition at all visits) for determination of CrCL. Blood pressure to be measured after resting in a semi-supine position for at least 5 minutes.
- 6. From the time a subject consents to participate in ING200336 and administration of IP at Day 1, only SAEs assessed as related to study participation (e.g., study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication, will be recorded in the eCRF for ING200336. Only SAEs related to study participation or to a concomitantly administered GSK or ViiV product will be collected between obtaining informed consent and administration of IP at Day 1. Note: At the time of the Withdrawal visit in ING117172 if there is an ongoing, unresolved adverse event (AE) and/or serious adverse event (SAE) it will be left in ING117172 as

<sup>\*\*</sup>HIV-1 RNA, lymphocyte subset, and laboratory assessment (hematology, chemistry, and urinalysis including a dipstick) data collected at the ING117172 unscheduled or last visit within 28 days of learning of the pregnancy will be transferred to serve as screening data in this study. The ING117172 Withdrawal visit will serve as the ING200336 Day 1. Gravidity: Maternal history and pregnancy risk assessment may occur at either Screening or Day 1 visit.

unresolved and transcribed as medical history in ING200336. If the AE and/or SAE worsen after enrollment into ING200336 it will be recorded on the AE/SAE forms in ING200336.

- 7. Intensive PK visit: The PK evaluations should be scheduled for study visits at Weeks 18-26, Weeks 30-36 and 8-12 weeks postpartum. The DTG dose on serial PK sampling days is to be given with a light meal/snack PK should be scheduled so that witnessed dosing of DTG/ABC/3TC FDC is as close as possible to 24 hours (generally 22-26 hours) after the previous dosing. The PK visit should be re-scheduled if the subject took their morning dose prior to coming into the clinic on the PK sampling day. See SPM for additional details.
- 8. If feasible, a cord and maternal blood sample will also be collected at delivery and if possible within 30 minutes of each other.
- 9. Suicidality Questionnaire will be conducted q 12 weeks during the Continuation Phase. 10. HIV-1 RNA and lymphocyte to be drawn within 24 hours of delivery and on the day of the post-partum PK evaluation.
- 11. The PGx sample should be collected at Day 1 if not collected during participation in ING117172, however this sample may be collected at any time during the study.
- 12. Plasma samples for storage will be collected at each visit for possible future analyses (including but not limited to HIV-1 RNA genotypic and phenotypic analyses in confirmed cases of subject withdrawal, HIV-1 RNA levels, when samples are lost or arrive at the laboratory unevaluable, and immunological parameters.)
- 13. Only for subjects who continue DTG/ABC/3TC and are seen in the clinic every 12 weeks until DTG/ABC/3TC is commercially available locally. Note: after delivery, subjects must use one of the contraception methods to avoid a 'new' pregnancy
- 14. A Follow up visit may be conducted approximately 4 weeks after the last dose of study provided IP, and is required only if the subject has ongoing SAEs or non-serious AEs (as outlined in the SPM) at the last on study visit. The assessments performed should reflect what is considered medically necessary to assess the event(s).

### 11.2. Appendix 2: Assessment Windows

Laboratory data and vital signs will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

A window around a target Study Day will typically include all days from the midpoints between it and the target Study Days of the previous and the proceeding visits. In general, the nominal target study day for week w is (7\*w)+1.

#### 11.2.1. Definitions of Assessment Windows for Analyses

| Analysis Set | Parameter | Target | Analysis | Analysis | |
|---|---|---|---|---|---|
| / Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| All | All | | | | Screening |
| | | 1 | | | Day 1 |
| | | 29 | 2 | 42 | Week 4 |
| | | 57 | 43 | 70 | Week 8 |
| | | 85 | 71 | 98 | Week 12 |
| | | 113 | 99 | 126 | Week 16 |
| | | 141 | 127 | 154 | Week 20 |
| | | 169 | 155 | 182 | Week 24 |
| | | 197 | 183 | 210 | Week 28 |
| | | 225 | 211 | 238 | Week 32 |
| | | 253 | 239 | 266 | Week 36 |
| | | 281 | 267 | 294 | Week 40 |
| | | 337 | 295 | 378 | Week 48 |
| | | 7*w+1 | 7*w-41 | 7*w+42 | Week w,<br>w=52, 64,<br>76, |
| | | Study Day of last dose<br>+ 28 | >Study Day<br>of last dose<br>+1 | >Study Day<br>of last dose<br>+1 | Follow-up |

#### NOTES:

- For parameters which are not scheduled to be assessed at particular visits, the all-inclusive windows defined will still be used.
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings.

# 11.2.2. Definitions of Assessment Windows for Inclusion in the PK Analysis

The windows for inclusion of PK samples in summary statistics for all PK visits will be as follows:

- Samples collected 15 minutes prior to dose for pre dose sample
- O Samples collected within ±15 min of the 1h and 2h time points
- o Samples collected within ± 30 min of the 3h, 4h, 6h time points
- o Samples collected within ± 1h for the 8h and 12h time points
- o Samples collected within ± 2h for the 24 h time point

#### 11.2.3. Stages of Pregnancy used for Pharmacokinetics

| Stage | | Weeks |
|-------------|-------------|-------|
| Ante-Partum | Trimester 2 | 18-26 |
| | Trimester 3 | 30-36 |
| Delivery | | |
| Post-Partum | | |

#### NOTES:

- Delivery is a single day.
- Post-partum PK assessment is done 8-12 weeks after delivery

#### 11.2.4. Analysis visits in relation to pregnancy

In addition, an analysis visit in relation to pregnancy is derived, which will also be listed in the listings.

- For the screening, delivery and post-partum visits, the same scheduled visit is used.
- For the Day 1 and ante-partum visits, the corresponding gestation weeks from reproductive system findings is used.
- For the subsequent post-partum visits, the analysis visit in relation to pregnancy is derived by (visit day of subsequent post-partum visit visit day at post-partum)/7.

## 11.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

### 11.3.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to Study Visits.

## 11.3.1.1. Treatment States for Laboratory, HIV Associated Conditions, Vital Signs, and Genotypic and Phenotypic Data

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date + 1 |

#### 11.3.1.2. Treatment States for Prior/Concomitant/Post-Therapy Medications Data

- Prior medications are those taken (i.e., started) before the start date of investigational product.
- Concomitant medications are those taken (i.e., started or continued) at any time between the start date and stop date of IP, inclusive. Prior medications that were continued during this period are also considered as concomitant medications.
- Post-treatment medications are those started after the stop date of IP.
   Concomitant medications that were continued during this period are also considered as post-treatment medications.

It will be assumed that medication has been taken on the date in which it is reported as started or stopped. Also, for any medication starting on the same date as IP, it will be assumed that the medication was taken after the subject started taking IP.

ART medications will also be classified as prior, concomitant and/or post-treatment according with the following modifications:

- ART starting on study treatment stop date will be considered as only posttreatment and not concomitant. It is expected that after discontinuation of study treatment, a subject may immediately begin taking another ART.
- ART stopping on study treatment start date will only be considered as prior and not concomitant.
- Any ART entered on the Prior ART eCRF with partial end date will be assumed to have finished before Screening.

| | Pre-<br>treatmen | t | On-tr | eatment | | Pos | st-treatm | ent | Prior | Conco-<br>mitant | Post |
|---|---|---|---|---|---|---|---|---|---|---|---|
| (a) | х х | | | | | | | | Υ | N | N |
| (b) | X | | | X | | | | | Υ | Υ | N |
| (c) | Х | | | | | | | X | Υ | Υ | Υ |
| (d) | | | X | X | | | | | N | Υ | N |
| (e) | | يو ا | X | | g. | Ŧ | | X | N | Υ | Υ |
| (f) | | IP Start Date | | | IP Stop Date | IP Stop Date+1 | X | X | N | N | Υ |
| (g) | ? x | ar l | | | do | p D | | | Υ | N | N |
| (h) | ? | Š | | X | St | Sto | | | Y* | Υ | N |
| (i) | ? | = | | | _ | ٩ | | X | Y* | Y* | Υ |
| (j) | x | | | | | | | ? | Υ | Y** | Y** |
| (k) | | | X | | | | | ? | N | Υ | Y** |
| (l) | | | | | | | X | ? | N | N | Υ |
| (m) | ? | | | | | | | ? | Y*** | Y*** | Y*** |
| (n) | x | X | | | | | | | Υ | Υ | N |
| (o) | ? | X | | | | | | | Y* | Y | N |
| (p) | ļ · | Х | | х | | | | | N | Υ | N |
| (p) | | X | | Α | Х | | | | N | Y | N |
| (r) | | | | | X | | | X | N | Υ | Υ |
| (s) | | | | | X | | | ? | N | Υ | Y** |
| (t) | | | | | | X | | X | N | N | Υ |
| (u) | | | | | | X | | ? | N | N | Υ |
| (v) | | | X | | | X | | | N | Υ | Υ |

x = start/stop date of medication

#### 11.3.1.3. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date |
| Onset Time Since<br>1st Dose (Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 |

<sup>? =</sup> missing start/stop date of medication

<sup>\*</sup> If a medication is stopped On-treatment or Post-treatment and no start date is recorded it will be assumed that the medication was ongoing from the Pre-treatment phase

<sup>\*\*</sup> If a medication is started Pre-treatment or On-treatment and no stop date is recorded then usage will be assumed to be ongoing for the remainder of the study

<sup>\*\*\*</sup> If a medication has no start or stop date it will be assumed that the medication was ongoing from the Pre-treatment phase to the Post-treatment phase

| Treatment State | Definition |
|-----------------|-----------------------------------------|
| | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on CRF. |

#### NOTES:

- In the case of a completely missing start date, the event will be considered to have started On-treatment unless
  an end date for the AE is provided which is before start of investigational product; in such a case the AE is
  assigned as Pre-treatment.
- If the IP Stop Date is missing, then any event with a start date on or after IP Start Date will be considered to be On-treatment.
  - If the start date of the AE is after IP Stop Date but has been recorded as potentially related to IP, then it will be classified as On-treatment.

#### 11.3.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Emergent | Emergent refers to AE Severity/ Lab toxicity that develops or increases in intensity after baseline |

#### NOTES:

- If the study treatment stop date is missing, then the AE/ Lab toxicity will be considered to be
  On-Treatment unless an end date for the AE/ Lab toxicity is provided which is before start of
  investigational product; in such a case the AE/ Lab toxicity is assigned as Pre-treatment.
- Time of study treatment dosing and start/stop time of AEs/ Lab toxicity should be considered, if collected.

#### 11.4. Appendix 4: Data Display Standards & Handling Conventions

#### 11.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | Reporting Area |
| HARP Server | : uk1salx00175 |
| HARP Compound : \ARPROD\GSK2619619\ING200336\Documents\final 01(SAC) | |
| Analysis Datasets | |

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1 or above).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented as SDTM.

#### Generation of RTF Files

RTF files will be generated for all reporting efforts.

#### 11.4.2. Reporting Standards

#### General

The current GSK Statistical Display Standards in the GSK Standards Library (IDSL) will be applied for reporting, unless otherwise stated (Library Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK Statistical Display Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the GSK Standard Statistical Display Principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to GSK Standard Statistical Display Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

| Unscheduled Visits | |
|---|---|
| <ul> <li>Unscheduled visit</li> </ul> | Unscheduled visits will be included in listings. |
| <ul> <li>Unscheduled visit</li> </ul> | s will be assigned to a study visit using the all-inclusive windows defined in Section |
| 11.2.1 | |
| Descriptive Summary | y Statistics |
| Continuous Data | Refer to GSK Standard Statistical Display Principle 6.06.1 |
| Categorical Data N, n, frequency, % | |
| Graphical Displays | |
| <ul> <li>Refer to GSK Standard Statistical Display Principals 7.01 to 7.13.</li> </ul> | |

### 11.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to Standards for the Transfer and Reporting of PK Data document. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to the GSK Standard PK Display Standard. Refer to the GSK Standard Statistical Display Principle 6.06.1. Note: If any concentration value is not calculable because of NQs, it will be excluded (set to missing) from the PK concentration Summary tables and Graphical displays and show as NQ in Listings. Refer to VQD-GUI-000722 (6.0) (Non-Compartmental Analysis of Pharmacokinetic Data) for handling of values below the Quantification Limit. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | The PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using WinNonLin v 5.2 or above. All calculations of non-compartmental parameters will be based on actual sampling times. |
| Pharmacokinetic Para | ameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | If any PK parameter is not calculable because of NQs, it will be excluded (set to missing) from the PK parameter summary. Refer to VQD-GUI-000722 (6.0) (Non-Compartmental Analysis of Pharmacokinetic Data) for handling of values below the Quantification Limit. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to GSK Standard PK Display Standard. |
| Untransformed PK parameter | tmax (TMAX), t1/2 |

#### 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

#### Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 11.2.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from initial study treatment start date:
  - Ref Date = Missing 
    → Study Day = Missing
  - Ref Date < Treatment Start Date → Study Day = Ref Date -Treatment Start Date
  - Ref Data ≥ Treatment Start Date → Study Day = Ref Date (Treatment Start Date) +
  - Note that Treatment Start Date is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### **Post Baseline**

Post-baseline refers to the combined time periods of On-treatment and Post-treatment.
 Post-baseline may be further specified according to phase of the study: Antepartum,
 Delivery, Postpartum or Continuation.

#### 11.5.2. Study Population

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
- Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:
- Cumulative Dose = Sum of (Number of Days x Total Daily Dose)
- If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Since only year of birth is recorded for subjects (day and month are not recorded), for the purpose of calculating age, day and month of birth will be imputed as '30th June'.

#### 11.5.3. Efficacy

#### **HIV-1 RNA**

Plasma for quantitative HIV-1 RNA will be collected. Methods to be used may include but
are not limited to the Abbott RealTime HIV-1 Assay lower limit of detection (LLOD) 40 c/mL.
In some cases (e.g., where the HIV-1 RNA is below the LLOD for a given assay) additional
exploratory methods may be used to further characterize HIV-1 RNA levels.

#### Lymphocyte

#### CD4+ Cell Count

Absolute CD4+ lymphocyte counts will be collected for assessment by flow cytometry.

#### 11.5.4. Safety

#### **Adverse Events**

#### AE Severity – DAIDS Grading.

- The DAIDS grading for severity of clinical adverse events will be performed.
- See protocol for DAIDS grading criteria.

#### **Suicidality Monitoring**

 Treatment emergent assessment of suicidality will be monitored during this study using the Columbia Suicide-Severity Rating Scale.

#### **Laboratory Parameters**

#### Lab Toxicities – DAIDS Grading

- The DAIDS grading for severity of clinical adverse events will be performed.
- See protocol for DAIDS grading criteria

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</li>

### 11.5.5. Pharmacokinetic

### PK Parameters

- The PK Population will include all subjects who undergo PK sampling and have evaluable PK assay results.
- See Table 5 for derived Pharmacokinetic parameters

### 11.6. Appendix 6: Reporting Standards for Missing Data

### 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as: Subjects are considered to have completed the study after completing the postpartum evaluation.</li> <li>Withdrawn participants were not replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables, listings and figures, unless otherwise specified.</li> </ul> |

### 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields<br/>on the collection instrument:</li> </ul> |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | <ul> <li>Any participants excluded from the summaries and/or statistical analyses will be<br/>documented along with the reason for exclusion in the clinical study report.</li> </ul> |

### 11.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in participant listing displays.</li> </ul> |
| Adverse<br>Events | <ul> <li>Imputations in the adverse events dataset are used for slotting events to the appropriate study time periods and for sorting in data listings.</li> <li>Partial dates for AE recorded in the CRF will be imputed using the following conventions:</li> </ul> |
| | If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month. Else if study treatment start date is not missing: If month and year of start date = month and year of study treatment start date then If stop date contains a full date and stop date is earlier than study treatment start date then set start date = 1st of month. Else set start date = study treatment start date. Else set start date = 1st of month. |
| | <ul> <li>Missing start day and month</li> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> </ul> </li> </ul> |

| Element | Reporting Detail | |
|---|---|---|
| | Missing stop day Missing stop day and month Completely missing start/end date | If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1. Else set start date = study treatment start date. Else set start date = January 1. Last day of the month will be used. No Imputation No imputation |
| | · | ng start or end dates will remain missing, with no imputation applied. |
| Concomitant<br>Medications/<br>Medical | | for any concomitant medications recorded in the CRF will be imputed lowing convention: |
| History | Missing start day | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing end day | A '28/29/30/31' will be used for the day (dependent on the month and year) |
| | Missing end day and month | A '31' will be used for the day and 'Dec' will be used for the month. |
| | Completely missing start/end date | No imputation |
| | The recorde | d partial date will be displayed in listings. |

### 11.7. Appendix 7: Values of Potential Clinical Importance

### 11.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Homotoprit | Ratio of | | | 0.54 |
| Hematocrit | 1 | $\Delta$ from BL | -0.075 | |
| Haamadahin | g/L | | | 180 |
| Haemoglobin | | $\Delta$ from BL | -25 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | <30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | <0.5 | >1.23 |
| Phosphorus | mmol/L | | <0.8 | >1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | <18 | >32 |

### 11.7.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >160 |
| Diastolic Blood Pressure | mmHg | <45 | >100 |
| Heart Rate | bpm | <40 | >110 |

### 11.8. Appendix 8: Abbreviations & Trademarks

### 11.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ABC | Abacavir |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AGA | Appropriate for Gestational Age |
| A&R | Analysis and Reporting |
| APGAR | Appearance, Pulse rate, Grimace, Activity, Respiration |
| CDISC | Clinical Data Interchange Standards Consortium |
| CD4+ | Helper-inducer T-lymphocyte having surface antigen CD4 (cluster of differentiation 4) |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CSR | Clinical Study Report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| DAIDS | Division of AIDS |
| DBF | Database Freeze |
| DBR | Database Release |
| DTG | Dolutegravir |
| eCRF | Electronic Case Record Form |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FDC | Fixed Dose Combination |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library (GSK Standards Library) |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT(E) | Intent-To-Treat (Exposed) |
| IUGR | Intrauterine Growth Restriction |
| LGA | Large for Gestational Age |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| RAP | Reporting & Analysis Plan |
| RNA | Ribonucleic acid |
| SAC | Statistical Analysis Complete |
| SAS | Statistical Analysis Software |
| SDTM | Study Data Tabulation Model |
| SGA | Small for Gestational Age |

### 11.8.2. Trademarks

| Trademarks of the ViiV Healthcare | Trademarks not owned by the ViiV<br>Healthcare |
|---|---|
| Dolutegravir | SAS |
| Epzicom/Kivexa | WinNonlin |

### 11.9. Appendix 9: List of Data Displays

All data displays will use the term "subject" rather than "participant" in accordance with CDSIC and GSK Statistical Display Standards.

#### 11.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|--------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | NA |
| Efficacy | 2.1 to 2.n | NA |
| Safety | 3.1 to 3.n | NA |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Virology | 5.1 | NA |
| Maternal and Infant Assessment | 6.1 to 6.n | NA |
| Section | Listi | ngs |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

### 11.9.2. Mock Example Shell Referencing

Nonstandard specifications will be referenced as indicated and if required example mockup displays provided in Appendix 9: Example Mock Shells for Data Displays.

| Section | Table | Listing |
|-------------------|--------|---------|
| Pharmacokinetic | PK Tn | PK Ln |
| Maternal Outcomes | MAT Tn | MAT Ln |
| Infant Outcomes | INF Tn | INF Ln |
| Virology | VIR Tn | NA |

NOTES: For displays having Example shell as \*, refer to TANGO Study (Compound: GSK3515864, Study ID: 204862, Reporting Effort: primary 01)

#### 11.9.3. Deliverables

| Delivery [Priority] | Description |
|---------------------|------------------------------------------------|
| IA SAC | Interim Analysis Statistical Analysis Complete |

## 11.9.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | ITT-E | ES1 | Summary of Subject Disposition for the Subject Conclusion Record overall and by relationship to COVID-19 Pandemic | Table will be summarised overall and then by COVID-19 relationship | IA SAC |
| 1.2. | Enrolled | NS3 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | IA SAC |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1.3. | ITT-E | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | IA SAC |
| 1.4. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | IA SAC |
| 1.5. | ITT-E | DM6 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | IA SAC |

### 11.9.5. Efficacy Tables

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Plasma | Plasma HIV-1 RNA | | | | |
| 2.1 | ITT-E | * | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit | | IA SAC |
| 2.2 | ITT-E | * | Proportion of Subjects with Plasma HIV-1 RNA <400 c/mL by Visit | | IA SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3 | ITT-E | * | Summary of Change from Baseline in HIV-1 RNA (c/mL) by Visit | | IA SAC |
| CD4+ C | ell Count | | | | |
| 2.4 | ITT-E | * | Summary of Change from Baseline in CD4+ Cell Count (cells/mm^3) by Visit | | IA SAC |
| Post- B | Post- Baseline Disease Progression | | | | |
| 2.5 | ITT-E | * | Summary of Post-Baseline HIV-1 Disease Progressions | | IA SAC |

### 11.9.6. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE5B | Summary of All Adverse Events by System Organ Class,<br>Preferred term and Maximum Toxicity | Ct.gov | IA SAC |
| 3.2. | Safety | AE3 | Summary of Grade 2-4 Adverse Events by Overall Frequency | ICH E3 | IA SAC |

| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.3. | Safety | AE15 | Summary of Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT | IA SAC |
| 3.4. | Safety | AE3 | Summary of Non-Serious Drug-Related Adverse Events by Overall Frequency | Plain Language Summary requirements (PLS). | IA SAC |
| 3.5. | Safety | AE16 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Number of Subjects and<br>Occurrences) | FDAAA, EudraCT | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.6. | Safety | AE20 | Summary of Serious Fatal and Non-Fatal Drug-Related Adverse by Overall Frequency | Plain Language Summary requirements (PLS). | IA SAC |
| 3.7. | Safety | AE8 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | | IA SAC |
| 3.8. | Safety | * | Summary of Maximum Post-Baseline Emergent Chemistry Toxicities | The key parameters would include ALT, AST, Total bilirubin, serum creatinine and GFR | IA SAC |
| 3.9. | Safety | * | Summary of Maximum Post-Baseline Emergent<br>Hematology Toxicities | The parameters would include<br>Hemoglobin, platelets, WBC | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit | The key parameters would include ALT, AST, Total bilirubin, serum creatinine and GFR | IA SAC |
| 3.11. | Safety | LB1 | Summary of Hematology Changes from Baseline by Visit | The parameters would include<br>Hemoglobin, platelets, WBC | IA SAC |
| 3.12. | Safety | LB1 | Summary of Urinalysis Changes from Baseline by Visit | Key parameters would be Urine protein/Creatinine ratio and Urine/Protein ratio | IA SAC |

ING200336

### 11.9.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| DTG PK | DTG PK | | | | |
| 4.1. | PK | PK01 | Summary of Plasma DTG PK Concentration-Time Data by Visit and Nominal Time Relative to Dose | | IA SAC |
| 4.2. | PK | PK T1 | Summary of untransformed and loge-transformed Derived Plasma DTG PK Parameters | | IA SAC |

### 11.9.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| DTG P | ( | | | | |
| 4.1. | PK | PK24 | Individual Plasma DTG Concentration-Time Plots (linear and Semi-log) | | IA SAC |
| 4.2. | PK | PK17 | Mean Plasma DTG Concentration-Time plots (linear and semilog) | | IA SAC |
| 4.3. | PK | PK18 | Median Plasma DTG Concentration-Time plots (linear and semi-log) | | IA SAC |

### 11.9.9. Virology Tables

| Virolog | Virology: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.1 | ITT-E | VIR T1 | Summary of Incidence of treatment-emergent genotypic and/or phenotypic resistance in subjects who meet confirmed virologic withdrawal criteria | | IA SAC |

ING200336

### 11.9.10. Maternal and Infant Assessment Tables

| Maternal ar | Maternal and Infant Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Standard/<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.1 | Safety | MAT T1 | Summary of Maternal Outcomes | | IA SAC |
| 6.2 | Safety | INF T1 | Summary of Infant Outcomes at Birth | | IA SAC |

## 11.9.11. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Standard /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | • | | | |
| 1. | ITT-E | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | IA SAC |
| Protoc | ol Deviations | | | | |
| 2. | ITT-E | DV2 | Listing of Important Protocol Deviations | ICH E3 | IA SAC |
| 3. | ITT-E | DV2 | Listing of all non-Important COVID-19 related Protocol Deviations | | IA SAC |
| Demog | raphic and Base | line Characterist | ics | | |
| 4. | ITT-E | DM2 | Listing of Demographic Characteristics | ICH E3 | IA SAC |
| 5. | ITT-E | DM9 | Listing of Race | ICH E3 | IA SAC |
| Exposi | ure and Treatmer | nt Compliance | | | |
| 6. | ITT-E | EX3 | Listing of Investigational Product Exposure Data | ICH E3 | IA SAC |
| Advers | e Events | | | | <u>.</u> |
| 7. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | IA SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Standard /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serious | s and Other Sign | ificant Adverse E | vents | | |
| 8. | Safety | AE8CPA | Listing of Non-Fatal Serious Adverse Events | ICH E3 | IA SAC |
| 9. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | IA SAC |
| 10. | Safety | AE8 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | ICH E3 | IA SAC |
| Labora | tory Assessment | ts | | | |
| 11. | Safety | LB5 | Listing of Clinical Chemistry Laboratory Data | ICH E3 | IA SAC |
| 12. | Safety | LB5 | Listing of Haematology Laboratory Data | ICH E3 | IA SAC |
| 13. | Safety | UR2 | Listing of Urinalysis Data | ICH E3 | IA SAC |

### 11.9.12. Non-ICH Listings

| Non-ICH: Listings | | | | |
|---|---|---|---|---|
| No. Population Example Shell Title Programming Notes Priority Programming Notes | | | | |
| Prior and | Concomitant | Medications | | |
| 14. | ITT-E | CM3 | Listing of Concomitant Medications | IA SAC |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 15. | ITT-E | CM3 | Listing of Prior ART Medications | Not Required | |
| 16. | ITT-E | CM3 | Listing of Concomitant ART Medications | | IA SAC |
| 17. | ITT-E | * | Listing of Relationship Between ATC Level 1, Ingredient and Verbatim Text | | IA SAC |
| 18. | ITT-E | * | Listing of Relationship Between ATC Level 4, Ingredient and Verbatim Text | | IA SAC |
| Adverse Events | | | | | |
| 19. | Safety | AE2 | Listing of Relationship Between Adverse Event System<br>Organ Classes, Preferred Terms, and Verbatim Text | | IA SAC |
| Pandemic | | | | | |
| 20. | Safety | PAN12 | Listing of COVID-19 Assessments and Symptom assessments | | IA SAC |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Non-Laboratory values | | | | | |
| 21. | Safety | ECSSRS4 | Listing of C-SSRS Suicidal Ideation and Behaviour Data | | IA SAC |
| Subject Disposition | | | | | |
| 22. | ITT-E | * | Listing of Investigational Product Accountability | | IA SAC |
| 23. | ITT-E | TA1 | Listing of Planned and Actual Treatments | | |
| 24. | All Subjects<br>Screened | * | Listing of Study Populations | | IA SAC |
| 25. | Enrolled | * | Listing of Subject Recruitment by Country and Site Number | Add a column "ARIA-ING117172<br>Unique Subject ID" | IA SAC |
| 26. | ITT-E | * | Listing of Visit Dates | | IA SAC |
| 27. | ITT-E | CDC3 | Listing of CDC Classification of HIV Infection at Baseline | | IA SAC |
| 28. | ITT-E | RF2 | Listing of HIV Risk Factors | | IA SAC |
| Medical Conditions | | | | | |
| 29. | ITT-E | MH2 | Listing of Current and Past Medical Conditions at Baseline | | IA SAC |
| Baseline ( | Characteristics | S | | | |
| 30. | ITT-E | * | Listing of Baseline Cardiovascular Risk Assessment Data | | IA SAC |
| 31. | ITT-E | * | Listing of History of Cardiac Therapeutic Procedures | | IA SAC |
| 32. | ITT-E | * | Listing of Cardiovascular Events at Baseline | | IA SAC |
| 33. | ITT-E | MAT L2 | Listing of Maternal History | | IA SAC |
| Efficacy | | | | | |
| 34. | ITT-E | * | Listing of Quantitative Plasma HIV-1 RNA | | IA SAC |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 35. | ITT-E | * | Listing of CD4+ Cell Count Data | | IA SAC |
| Vital Signs | | | | | |
| 36. | Safety | VS4 | Listing of All Vital Signs Data | | IA SAC |
| PK Endpoints | | | | | |
| 37. | PK | PK L1 | Listing of Plasma DTG PK Concentration-Time Data | | IA SAC |
| 38. | PK | PK L2 | Listing of Plasma DTG PK Parameters | | IA SAC |
| Maternal and Infant Endpoints | | | | | |
| 39. | Safety | MAT L1 | Listing of Maternal Outcomes | | IA SAC |
| 40. | Safety | MAT L3 | Listing of Pregnancy Risk Assessment | | IA SAC |
| 41. | Safety | INF L1 | Listing of Infant Outcomes | | IA SAC |

### 11.10. Appendix 10: Example Mock Shells for Data Displays

Example mock shells for Data Displays will be provided in a separate document.